## Statistical Analysis Plan

Protocol Title: A Prospective, Multi-Center, Open Label, Single Arm Clinical Trial Evaluating the Safety and Efficacy of the Cordella™ Pulmonary Artery Sensor System in New York Heart Association (NYHA) Class III Heart Failure Patients

Brief Title: PROACTIVE-HF IDE Trial Heart Failure NYHA Class III

Unique Protocol ID: ETX-HFS-PA-03

NCT04089059

17 Aug 2023

## **Statistical Analysis Plan**

**Sponsor Name:** Endotronix

**Protocol Number:** ETX-HFS-PA-03

Protocol Title: A <u>Pro</u>spective, Multi-Center, Open L<u>a</u>bel, Single Arm Clinical <u>Tri</u>al E<u>v</u>aluating the Safety and <u>E</u>fficacy of the Cordella <sup>™</sup> Pulmonary Artery Sensor System in New York Heart Association (NYHA) Class III <u>H</u>eart <u>F</u>ailure Patients

(PROACTIVE- HF Trial)

Investigational Product Name: Cordella Pulmonary Artery Sensor System
Protocol Version and Date: Version 10.0 dated 16 Dec 2022

IDE Number: G190020

Syneos Health Project Code: 7000235

Author: Stone Liu, Biostatistician I

Version: 3.0 Dated: 17 Aug 2023

#### **Notice of Confidential and Proprietary Information:**

The information contained in this document is confidential belonging to Endotronix. Acceptance of this document constitutes agreement by the recipient that no information contained herein will be published or disclosed without prior written authorization from an official of Endotronix. However, this document may be disclosed to appropriate Institutional Review Board and Ethics Committees or duly authorized representatives of a national regulatory authority under the condition that they are requested to keep it confidential. In the event of an actual or suspected breach of this obligation, Syneos Health should be notified promptly.

## **Revision History**

| Version # | Date<br>(DD-Mmm-YYYY) | Document Owner | Revision Summary |
|---|---|---|---|
| 1.0 | 22-Jun-2020 | Natalie Steigerwald | Initial Release Version |
| 2.0 | 29-Dec-2022 | Stone Liu | Updated according to protocol V9.0 |
| | | | Repeated the primary safety analysis on ITT additionally. The cutoff for 6 month analysis updated to 180 days from 183 days Added an AE summary for 'Other serious adverse events (AE) CEC adjudicated' |
| | | Stone Liu | Added separate analyses of HFH and all-cause mortality from CEC adjudication results The compression population update to Cohort #1, Cohort #2 and #3 from Cohort #1 and Cohort #2 |
| 2.1 | 17-Aug-2023 | | The secondary endpoint #3 update to Comparison of the number of HF Hospitalizations or Emergency Department/ Hospital Outpatient IV diuretic visits of Cohort #1 and Cohort #2 + #3 at 6 and 12 months post implant from Comparison of the number of HF Hospitalizations or Emergency Department/ Hospital Outpatient IV diuretic visits of Cohort #1 and Cohort #2 at 6 and 12 months post implant |
| | | | The secondary endpoint #14 Change from baseline in PAP parameters collected via CorPASS will not performed for Cohort #1 population |

I confirm that I have reviewed this document and agree with the content.

| Approvals | | |
|---|---|---|
| Syneos Health Approval | | |
| Stone Liu, Biostatistician I | Store Liu | Electronically signed by: Stone Liu<br>Reason: I am the author<br>Date: Aug 17, 2023 14:58 GMT+8 |
| Lead Biostatistician | Signature | Date (DD-Mmm-YYYY) |
| Wesley Basson, Principal Stat Programmer | Wesley Basson | Electronically signed by: Wesley Basson<br>Reason: I am the approver<br>Date: Aug 17, 2023 10:28 GMT+2 |
| Lead Statistical Programmer | Signature | Date (DD-Mmm-YYYY) |
| Tianzhe Liu, Assoc Dir, Biostatistics | Tenz lu | Electronically signed by: Tianzhe Liu<br>Reason: I am the reviewer<br>Date: Aug 17, 2023 17:52 GMT+8 |
| Senior Reviewing Biostatistician | Signature | Date (DD-Mmm-YYYY) |
| _ | | |
| En | dotronix, Inc. | |
| Andrea Sauerland, Vice President Clinical Operations | Andrea Sauerland | Electronically signed by: Andrea<br>Sauerland<br>Reason: I am the approver<br>Date: Aug 17, 2023 09:11 GMT+2 |
| Sponsor Contact | Signature | Date (DD-Mmm-YYYY) |

## **Table of Contents**

| Rev | ision H | istory | 2 |
|---|---|---|---|
| Арр | orovals | | 3 |
| 1. | Purpo | ose | 11 |
| | 1.1. | Responsibilities | 11 |
| | 1.2. | Timings of Analyses | 11 |
| 2. | Study | / Objectives | 12 |
| | 2.1. | Study Objective | 12 |
| | 2.2. | Brief Description | 12 |
| | 2.3. | Subject Selection | 15 |
| | | 2.3.1. Inclusion Criteria | 15 |
| | | 2.3.2. Exclusion Criteria | 15 |
| | 2.4. | Determination of Sample Size | 16 |
| | | 2.4.1. Primary Efficacy Endpoint (at 6 months post- implant) | 16 |
| | | 2.4.2. Additional Secondary Efficacy Endpoints | 19 |
| | | 2.4.3. Primary Safety Endpoints | 20 |
| | 2.5. | Treatment Assignment & Blinding | 21 |
| | 2.6. | Study Device | 21 |
| | 2.7. | Study Procedures and Time and Event Schedule | 22 |
| 3. | Endp | oints | 23 |
| | 3.1. | Primary Efficacy Endpoint | 23 |
| | 3.2. | Primary Safety Endpoints | 23 |
| | 3.3. | Secondary Efficacy Endpoints | 23 |
| | 3.4. | Secondary Safety Endpoints | 24 |
| 4. | Analy | rsis Sets | 25 |
| | 4.1. | Enrolled Set. | 25 |
| | 4.2. | Intent-to-Treat Population | 25 |
| | 4.3. | Modified Intent-to-Treat Population (mITT) | 25 |
| | 4.4. | Per Protocol Population | 25 |
| | 4.5. | Cohort #1 Population | 25 |
| | 4.6. | Comparison Population | 25 |
| | 4.7. | Protocol Deviations | 25 |

| 5. | Gene | ral Aspec | ts for Statistical Analysis | 26 |
|---|---|---|---|---|
| | 5.1. | Genera | ll Methods | 26 |
| | 5.2. | Key De | finitions | 26 |
| | 5.3. | Missing Data | | |
| | 5.4. | Visit Wi | indows | 27 |
| | 5.5. | Pooling | of Sites | 27 |
| | 5.6. | Subgro | ups | 28 |
| 6. | Demo | ographic, | Other Baseline Characteristics and Medication | 29 |
| | 6.1. | Subject | t Disposition and Withdrawals | 29 |
| | 6.2. | Demog | raphic | 29 |
| | 6.3. | Medica | l History and Concomitant Diseases | 29 |
| | 6.4. | Other B | Baseline Characteristics | 29 |
| | 6.5. | Medica | tion | 29 |
| | | 6.5.1. | Baseline Medication | 29 |
| | | 6.5.2. | Concomitant Medication | 30 |
| 7. | Effica | юу | | 31 |
| | 7.1. | Primary | Efficacy Endpoint and Analysis | 31 |
| | | 7.1.1. | Main analysis | 31 |
| | | 7.1.2. | Sensitivity analysis | 31 |
| | | 7.1.3. | Supplementary analysis | 32 |
| | | 7.1.4. | Incidence of HF Hospitalizations or all-cause mortality at 12 months | 32 |
| | | 7.1.5. | Number of HF Hospitalizations at 6 and 12 months post-implant compare number of HF Hospitalizations in the 6 and 12 months prior to implant | |
| | | 7.1.6. | Comparison of the number of HF Hospitalizations or Emergency Dep<br>Hospital Outpatient IV diuretic visits of Cohort #1 and Cohort #2 + Cohor<br>and 12 month post implant | rt #3 at 6 |
| | | 7.1.7. | Change of NT-proBNP from Baseline through 6 and 12 months | 33 |
| | | 7.1.8. | Combined outcome of: a. First and recurrent HF Hospitalizations b. Emergency Department/ Hospital Outpatient IV diuretic visits c. all-cause at 6 months | mortality |
| | | 7.1.9. | Heart failure hospitalization or HF Emergency Department / Hospital Out diuretic visits at 6 and 12 months | • |
| | | 7.1.10. | Cardiac and all-cause mortality | 34 |
| | | 7.1.11. | Days Alive and Out of Hospital (DAOH) | 35 |

| | | 7.1.12. | Hospital Outpatient IV diuretic visits | 35 |
|---|---|---|---|---|
| | | 7.1.13. | Heart failure related medication changes | 35 |
| | | 7.1.14. | Change in PA pressure | 35 |
| | | 7.1.15. | Percentage of device success as documented by ability of the System successfully transmit PAP data | |
| | | 7.1.16. | Subject Outcome Measures, measured by Quality of Life KCCQ questionnain | re36 |
| | | 7.1.17. | Functional status improvement measured by NYHA and 6-Minute Walk Test | 36 |
| 8. | Safety | y | | 38 |
| | 8.1. | Primary | safety endpoint | 38 |
| | | 8.1.1. | Main analysis | 38 |
| | | 8.1.2. | Sensitivity analysis | 38 |
| | 8.2. | Second | ary safety endpoints | 39 |
| | 8.3. | Adverse | e Events | 39 |
| | | 8.3.2. | Relationship | 39 |
| | | 8.3.3. | Predefined AE categories | 40 |
| | | 8.3.4. | Presentation | 40 |
| | 8.4. | Laborat | ory Evaluations | 42 |
| | 8.5. | Vital Sig | gns | 43 |
| | 8.6. | Electro | cardiogram (ECG) | 43 |
| | 8.7. | Echoca | rdiogram | 43 |
| | 8.8. | Physica | ll Examination | 44 |
| 9. | Interir | m Analyse | es | 45 |
| 10. | Chan | ges from | Analysis Planned in Protocol | 46 |
| 11. | | | ······································ | |
| 12. | Progr | amming ( | Considerations | 48 |
| | 12.1. | Genera | l Considerations | 48 |
| | 12.2. | Table, I | _isting, and Figure Format | 48 |
| | | 12.2.1. | General | 48 |
| | | 12.2.2. | Headers | 48 |
| | | 12.2.3. | Display Titles | 49 |
| | | 12.2.4. | Body of the Data Display | 49 |
| | | 12.2.5. | Footnotes | 50 |
| 13. | Qualit | y Control | | 51 |

# **Statistical Analysis Plan for Interventional Studies** Sponsor: Endotronix, Protocol No.: ETX-HFS-PA-03

| 14. | Index of Tables | . 52 |
|---|---|---|
| 15. | Index of Figures | . 73 |
| 16. | Index of Listings | . 77 |
| 17. | Appendices | . 80 |
| | 17.1. Appendix 1: Time and Event Schedule | .81 |
| | 17.2. Appendix 2: The Kansas City Cardiomyopathy Questionnaire Scoring Instruction | ons |
| | | . 82 |

## Glossary of Abbreviations

| Abbreviation | Description |
|---|---|
| ACC | American College of Cardiology |
| ACE-I | Angiotensin Converting Enzyme-Inhibitors |
| ADE | Adverse Device Effect |
| AE | Adverse Event |
| AHA | American Heart Association |
| ALT | Alanine Aminotransferase |
| ARB | Angiotensin Receptor Blockers |
| ARNI | Angiotensin-Neprilysin Inhibitors |
| ATC | Anatomical Therapeutic Chemical |
| AST | Aspartate Aminotransferase |
| ВМІ | Body Mass index |
| BNP | Brain Natriuretic Peptide |
| BP | Blood Pressure |
| BUN | Blood Urea Nitrogen |
| CalEQ | Cordella™ Calibration Equipment |
| CDAP | Cordella Data Analysis Platform |
| CE | Conformité Européene/European Conformity |
| CI | Confidence Interval |
| CDAP | CorPASS Data Analysis Platform |
| Cordella System | Cordella™ Heart Failure System |
| cm | Centimeters |
| CorPASS | Cordella™ Pulmonary Artery Sensor System |
| CRO | Contract Research Organization |
| CRP | C- Reactive Protein |
| CRT | Cardiac Resynchronization Therapy |
| CRT-D | Cardiac Resynchronization Therapy Defibrillator |
| CRT-P | Cardiac Resynchronization Therapy Pacemaker P |
| CS | Clinically Significant |
| CV | Cardiovascular |
| eCRF | Electronic Case Report Form |

| Abbreviation | Description |
|--------------|------------------------------------------------|
| DD | Device Deficiency |
| dPAP | Diastolic Pulmonary Artery Pressure |
| DSMB | Data Safety Monitoring Board |
| DSRC | Device/System Related Complication |
| ED | Emergency Department |
| ECG | Electrocardiogram |
| GDMT | Guideline Directed Medical Therapy |
| GFR | Glomerular Filtration Rate |
| HF | Heart Failure |
| HFH | Heart Failure Hospitalization |
| HFEF | Heart Failure Ejection Fraction |
| HFpEF | Heart Failure with Preserved Ejection Fraction |
| HFrEF | Heart Failure with Reduced Ejection Fraction |
| HR | Heart Rate |
| INR | International Normalized Ratio |
| ІТТ | Intent to Treat |
| IWRS | Interactive Web Response System |
| KCCQ | Kansas City Cardiomyopathy Questionnaire |
| lb | Pound |
| LVEDD | Left Ventricular End Diastolic Dimension |
| LVEF | Left Ventricular Ejection Fraction |
| MAR | Missing at Random |
| Max | Maximum |
| MedDRA | Medical Dictionary for Regulatory Activities |
| Min | Minimum |
| mITT | Modified Intent to Treat |
| MNAR | Missing not at Random |
| mPAP | Mean Pulmonary Artery Pressure |
| N/A | Not Applicable |
| NCS | Not Clinically Significant |
| NYHA | New York Heart Association |

| Abbreviation | Description |
|--------------|-----------------------------------------|
| PT | Preferred Term |
| PAP | Pulmonary Artery Pressure |
| PCWP | Pulmonary Capillary Wedge Pressure |
| рН | Potential of Hydrogen |
| PMA | Premarket Approval |
| PMP | myCordella™ Patient Management Portal |
| PP | Per protocol |
| PTT | Partial Thromboplastin Time |
| QC | Quality Control |
| QTc | Corrected QT Interval |
| RAP | Right Atrial Pressure |
| RBC | Red Blood Cell |
| RHC | Right Heart Catheterization |
| RVP | Right Ventricular Pressure |
| SAE | Serious Adverse Event |
| SADE | Serious Adverse Device Effects |
| SAP | Statistical Analysis Plan |
| SD | Standard Deviation |
| SI | Standard International System of Units |
| SGOT | Serum Glutamic Oxaloacetic Transaminase |
| SGPT | Serum Glutamic Pyruvic Transaminase |
| SpO2 | Peripheral capillary oxygen saturation |
| sPAP | Systolic Pulmonary Artery Pressure |
| SOC | System Organ Class |
| SOP | Standard Operating Procedure |
| TFL | Table, Figure and Listing |
| WHO | World Health Organization |
| UADE | Unanticipated Adverse Device Effect |

### 1. Purpose

The purpose of this statistical analysis plan (SAP) is to ensure that the data listings, summary tables and figures which will be produced, and the statistical methodologies that will be used, are complete and appropriate to allow valid conclusions regarding the study objectives.

## 1.1. Responsibilities

Syneos Health will perform the statistical analyses and is responsible for the production and quality control of all tables, figures, and listings. Health Economic analysis will be covered in a separate SAP.

Assessment of protocol deviations as minor or major for the definition of the analysis sets remains with the Sponsor.

#### 1.2. Timings of Analyses

Main analysis will be performed after all Cohort #2-Previously enrolled Treatment Arm subjects and Cohort #3- Newly enrolled subjects completed the Month 6(V5) study visit or discontinued earlier. This main analysis will include all endpoints and analyses described in the SAP as far as data allow. The cleaning process will be completed at this stage, saying that the main analysis will be based on clean and coded data. Protocol deviations will be assessed and analysis sets will be defined following Syneos Health SOP (Blind) Data Review and Definition of Analysis Sets (3911) prior to the cut-off date for database (soft) lock. At this stage it will be decided if the analysis based on the Per-protocol population will be performed. Analysis will be performed on all analysis sets deemed relevant for the analysis. Listings will include all data collected until the cut-off date, by visit summaries will include data until V5 (Month 6), summaries (e.g. medication, or adverse events) without visit information will include all data until the cut-off date.

Additionally, an analysis on safety data will be performed once, the first 50 subjects which have been implanted with the Cordella PA Sensor have completed V4, Month 3 and also when 100 subjects have completed V3, Month 1. These safety analyses may occur at the same time depending on the timing of study visits. Analysis will be done on as much as possible clean and coded safety data.

The follow-up (final) analysis is planned after all subjects have completed the final study visit (V9, Year 3) or terminated early from the study.

An independent Data Safety Monitoring Board (DSMB) will review descriptive summaries of accumulating safety and subject disposition data on regular basis. Further description of the DSMB analyses can be found in the DSMB Statistical Analysis Plan Version 3.1 dated 07-Feb-2022 [1] and the DSMB charter Version 4.0 dated 04-Mar-2022 [1]. The study team from Syneos Health Biostatistics will perform the analyses.

The cut-off time point for the safety analysis and first two DSMB meetings expected to the identical. Outputs described in the DSMB SAP will cover the safety and DSMB analysis.

## 2. Study Objectives

#### 2.1. Study Objective

To demonstrate safety and efficacy of the Cordella PA Sensor System.

#### 2.2. Brief Description

This is a prospective, open-label, single arm, multi-center clinical trial evaluating the safety and efficacy of the Cordella™ Pulmonary Artery Sensor System in New York Heart Association (NYHA) Class III heart failure (HF) subjects compared to a Performance Goal (PG).

All eligible subjects get implanted the Cordella PA Sensor. As part of the Cordella PA Sensor System (CorPASS), it intends to measure, record, and transmit pulmonary artery pressure (PAP) data from NYHA Class III heart failure patients at home to clinicians for assessment and patient-centered HF management, with the goal of reducing heart failure hospitalizations.

The study is planned to be conducted in up to 120 sites in the United States and Europe. The study population includes male and female subjects, ≥ 18 years of age with a diagnosis of NYHA Class III heart failure.

With this amendment to the protocol/CIP, subjects will be categorized into three (3) different cohorts:

- 1. Cohort #1- Previously enrolled Control Arm subjects
  - Subjects in this cohort will be unblinded to their PAP measurements and informed about their previous group assignment and continue their Follow-up visit schedule
  - Additionally, subjects will be asked, throughout the remaining Follow-up period, to complete a regular subject survey on their experience with PAP Measurements and PAP Values.
  - Clinicians will be unblinded to their PAP measurements and start managing the patients to target PA pressures per protocol/ CIP and according to Guideline Directed Medical Therapy (GDMT)
  - Additionally, the clinical site will be asked to contact the subject on a regular basis to discuss their PAP values
  - Separate analysis (safety and effectiveness) will be performed for Cohort #1
- 2. Cohort #2- Previously enrolled Treatment Arm subjects
  - As of month 12 subjects in this cohort will be able to see their own PAP measurements for the remaining duration of the study.
  - Clinicians will continue to manage the patients to target PA pressures per protocol/CIP and according to GDMT
  - All primary and secondary safety and effectiveness analyses will be performed
- 3. Cohort #3- Newly enrolled subjects

- Subjects will participate in the Screening/ Enrollment Visit, Cordella PA Sensor Implant Visit, and Follow-Up Visits.
- Clinicians will manage the patients to target PA pressures per protocol/ CIP and according to GDMT.
- As of month 12 subjects in this cohort will be able to see their own PAP measurements for the remaining duration of the study.
- All primary and secondary safety and effectiveness analyses will be performed.

Up to 450 subjects are planned to be enrolled and successfully implanted with the Cordella PA (consisting of subjects from Cohort #2 and Cohort #3 below). These subjects will be the basis for the primary study analysis. Additionally, up to 85 subjects (cross- over from former Control Arm) will continued to be followed in Cohort #1.

To be enrolled into the study, subjects must be receiving stable Guideline Directed Medical Therapy (GDMT) for HF per current American Heart Association (AHA)/American College of Cardiology (ACC) guidelines as standard-of-care for HF therapy in the United States and Europe, with any intolerance documented for at least 30 days. This will be verified by the trial specific PROACTIVE-HF Clinical Eligibility Committee.

Subjects must be diagnosed with heart failure for a minimum of 3 months, are clinically stable, have an increase of NT-proBNP and a HF related hospitalization, HF treatment in a hospital day-care setting, or urgent outpatient clinic HF visit for IV diuretics within 12 month (last hospitalization should be 30 days before Screening /Enrollment)

Potential subjects are to be identified by the Investigator and research staff with the study Inclusion and Exclusion criteria in mind. At Screening, subjects are fully informed on what to expect with study participation to maintain a high study participation retention rate. As part of the study Implant Visit, subjects undergo a training on the at-home use of the Cordella™ Heart Failure System (Cordella System) to ensure compliance with the web-based clinical care management component of the Cordella™ Heart Failure System. Throughout the study, subjects will continue to be followed closely to ensure study compliance as well as continued study participation

At the Screening/Enrollment Visit, subjects review and sign the informed consent form prior to any study-related procedures performed. Based on Screening Visit results, the Investigator confirms and documents study eligibility for each subject. As part of the study screening process, subjects will be scheduled for a RHC and PA Sensor Implant procedure.

At the Implant Visit (V2), the Cordella PA Sensor, which is pre-mounted on a catheter Delivery System, is delivered according to the system's Instructions for Use. Once deployed, the Sensor PAP readings are calibrated using the system's fluid-filled catheter. The calibration coefficients for that Sensor/subject are stored in a database, allowing for consistent PAP calculations throughout the study duration.

Below enrollment stopping rules will be considered during the study.

- 1) to have sufficient number of women representatives in the study, it is anticipated to include at least 35 % women out of the planned population. Therefore, the inclusion/enrollment of the men subjects will be limited to 65% at the most.
- 2) to have sufficient number of heart failure with preserved ejection fraction (HFpEF) representatives in the study, it is anticipated to include at least 45 % HFpEF subjects out of the planned population.

Therefore, the inclusion/enrollment of the heart failure with reduced ejection fraction (HFrEF) subjects will be limited to 55% at the most.

Subjects are observed until stable and discharged home with instructions to take their PAP measurements daily (e.g. same time each morning) along with their weight, BP, HR and SpO2, which are wirelessly transmitted to a secure website. Subjects also receive a Cordella ™ PA Sensor System implant card, a Patient User's Manual, and a Technical Support number to contact Endotronix representatives with any questions.

The clinician will contact all subjects on a pre-determined call schedule basis to discuss their health status and all patients will be treated according to GDMT.

Visibility to patients' daily data trends will enable the clinician to proactively manage the patients to target PA pressures per protocol and according to GDMT.

Subjects return for follow up visits at 1, 6, 12, 18, 24 months and Year 3 after the Cordella PA Sensor implant, or until study termination. The 3-month follow-up visit will be performed as remote/ virtual Telemonitoring visit.

A subject may discontinue his or her participation without giving a reason at any time during the study. Should a subject's participation be discontinued, the primary reason for termination has to be recorded in the Electronic Case Report Form (eCRF). In addition, efforts have to be made to perform all procedures scheduled for the Month 6 (V5) visit if discontinuation is prior to that visit, or the year 3 (V9) visit if discontinuation is after year 2 but before Year 3. Subjects who are withdrawn may be replaced with new subjects for evaluation upon Sponsor approval.

The primary reason for discontinuation or withdrawal of the subject from the study is collected using the following categories:

- Lost to follow-up. The subject did not return to the clinic and attempts to contact the subject were unsuccessful.
- Voluntary withdrawal. The subject wishes to withdraw from the study. The reason for withdrawal, if provided, recorded in the eCRF.
- Principal Investigator withdrawal due to failure to comply with trial requirements or subject is uncooperative or refuses to continue in the trial
- Study termination. The sponsor, Institutional Review Board (IRB), or regulatory agency terminates the study
- Other

After completion of the last study visit (V9) the subject continues to participate in the site-specific Heart Failure Follow-up program.

Main analysis to demonstrate durability of the treatment effect is planned to be performed at the timepoint, when all Cohort #2 and #3 subjects have completed 6 months of follow-up or discontinued study earlier. At this timepoint the complete analysis as defined in the SAP will be performed, including definition of the protocol deviations and analysis sets. The analysis will be done on the clean and coded data.

Once all subjects completed the final study visit (V9) or terminated early from the study, a follow-up analysis will be done. For the follow-up analysis, the complete set of outputs will be refreshed based on the data available at study end.

DSMB meetings are planned for the study and will follow the scheduled defined in the DSMB charter.

#### 2.3. Subject Selection

Subjects in this study are male or female NYHA Class III heart failure patients at least 18 years of age. Subjects must be diagnosed with heart failure for a minimum of 3 months, are clinically stable, have an increase of NT-proBNP and a HF related hospitalization, HF treatment in a hospital day-care setting, or urgent outpatient clinic HF visit for IV diuretics within 12 months (last hospitalization should be 30 days before Screening /Enrollment). Subjects must also meet certain physical requirements necessary for the Cordella PA Sensor implant and functionality of the Cordella System as outlined in the study Inclusion/Exclusion Criteria below.

#### 2.3.1. Inclusion Criteria

In order to be eligible to participate in this study, each subject must meet all of the following criteria:

- 1. Subject has given written informed consent
- 2. Male or female, at least 18 years of age
- 3. Diagnosis and treatment of HF (regardless of left ventricular ejection fraction (LVEF)) for ≥ 3 months and NYHA Class III HF at time of Screening
- 4. Subjects should be on stable, optimally titrated medical therapy for at least 30 days, as recommended according to current American Heart Association (AHA)/American College of Cardiology (ACC) guidelines as standard-of-care for HF therapy in the United States, with any intolerance documented.
- 5. HF related hospitalization, HF treatment in a hospital day-care setting, or urgent outpatient clinic HF visit for IV diuretics within 12 month (last hospitalization should be 30 days before Screening /Enrollment) and/or N-terminal pro B-type Natriuretic Peptide (NTproBNP) at time of Screening/Enrollment defined as:
  - a. Subjects with LVEF ≤ 50%: NT-proBNP ≥ 1500 pg/mL.
  - b. Subjects with LVEF > 50%: NT-proBNP ≥ 800 pg/mL.

Thresholds for NT-proBNP (for both LVEF ≤ 50% and LVEF > 50%) will be corrected for body mass index (BMI) using a 4% reduction per BMI unit over 25 kg/m<sup>2</sup>

- 6. Subjects should be on diuretic therapy
- 7. Subjects who are physically able to hold the myCordella™ Patient Reader unit (approximate weight 1.3lb) against the ventral thoracic surface for up to 2 minutes per day while in a seated position, as well as dock and undock the myCordella™ Patient Reader
- 8. Subjects with sufficient eyesight, hearing, and mental capacity to respond to the myCordella™ Patient Reader's audio/visual cues and operate the myCordella™ Patient Reader
- 9. Subject has sufficient Cellular and/ or Wi- Fi Internet coverage at home
- 10. Subject agrees to return to the treating Investigator for all scheduled follow up visits and can return to the hospital for follow up

#### 2.3.2. Exclusion Criteria

A potential subject who meets any of the following criteria will be excluded from participation in this study:

1. Intolerance to all neuro-hormonal antagonists (i.e., intolerance to angiotensin converting enzyme-inhibitors (ACE-I), angiotensin receptor blockers (ARB), angiotensin-neprilysin inhibitors (ARNI), and beta-blockers) due to hypotension or renal dysfunction

This document is confidential.

SAP Version: 3.0 dated 17-Aug-2023

Controlled Document ID: 3903A.01, Effective Date 29-Oct-2018

- 2. ACC/AHA Stage D refractory HF (including having received or currently receiving pharmacologic circulatory support with inotropes)
- 3. Subjects with history of recurrent pulmonary embolism (≥ 2 episodes within 5 years prior to Screening Visit) and/or deep vein thrombosis within 3 months of the Screening Visit
- 4. Subjects who have had a major cardiovascular (CV) event (e.g., myocardial infarction, stroke) within 3 months of the Screening Visit
- 5. Unrepaired severe valvular disease
- 6. Subjects with significant congenital heart disease that has not been repaired and would prevent implantation of the Cordella PA Sensor or mechanical/tissue right heart valve(s)
- 7. Subjects with known coagulation disorders
- 8. Subjects with a hypersensitivity or allergy to platelet aggregation inhibitors including aspirin, clopidogrel, prasugrel, and ticagrelor; or patients unable to take dual antiplatelet or anticoagulants for one- month post implant
- 9. Known history of life threatening allergy to contrast dye.
- 10. Subjects whereby RHC is contraindicated
- 11. Subjects with an active infection at the Sensor Implant Visit
- 12. Subjects with a Glomerular Filtration Rate (GFR) < 25 ml/min or who are on chronic renal dialysis
- 13. Implanted with Cardiac Resynchronization Therapy (CRT) Pacemaker P (CRT-P) or CRT-Defibrillator (CRT-D) for less than 90 days prior to screening visit
- 14. Received or are likely to receive an advanced therapy (e.g., mechanical circulatory support or lung or heart transplant) in the next 12 months
- 15. Subjects who are pregnant or breastfeeding
- 16. Subjects who are unwilling or deemed by the Investigator to be unwilling to comply with the study protocol, or subjects with a history of non-compliance
- 17. Severe illness, other than heart disease, which would limit survival to <1 year
- 18. Subjects whose clinical condition, in the opinion of the Investigator, makes them an unsuitable candidate for the study
- 19. Subjects enrolled in another investigational trial with an active Treatment Arm
- 20. Subject who is in custody by order of an authority or a court of law

#### 2.4. Determination of Sample Size

2.4.1. Primary Efficacy Endpoint (at 6 months post- implant)

To meet the objectives of the study, observed event rates in the single arm PROACTIVE-HF should be similar to observed event rates in the treatment arm of CardioMEMS studies. Furthermore, observed event rates in the single arm PROACTIVE-HF should be lower than observed event rates in the control arm of CardioMEMS studies.

Thus, we set the performance goal (PG) as the LOWER of 1) the meta-analysis upper bound confidence interval of CardioMEMS treated patients, and 2) the meta-analysis estimates of CardioMEMS control patients, further adjusted down by potential impact of SGLT2i.

Furthermore, we also require that the single arm PROACTIVE-HF observed event rate is LOWER than both 1) the meta-analysis estimate of CardioMEMS treatment patients, and 2) the lowest observed event rates of CardioMEMS control patients, further adjusted down by potential impact of SGLT2i.

The primary endpoint will be the 6 month incidence of HF related Hospitalizations (HFH) or all-cause mortality compared to PG.

The endpoint PG is based on a random effects meta-analysis for the log-transformed incidence rate fit via restricted maximum likelihood. Results are back transformed to the rate scale. Calculations were performed in R version 3.6.3 with the "metafor" package.

The mean 6 month event rate from the meta-analysis of prior control studies is 0.46, or 0.43 on an adjusted basis to account for SGLT2i inclusion in the guidelines (Adjustment applied assuming 50% use of SGLT2i at the average hazard ratio observed across EMPEROR Preserved, EMPEROR REDUCED, DAPA-HF for NYHA III subjects.). A 6 month event rate of 0.43 also represents a value just below both the highest event rate observed across the CardioMEMS treatment studies (0.44 in MEMS-HF) and the upper bound of the overall meta-analytic treatment estimate (0.44). Taking the totality of results from the meta-analysis of active treatment trials, individual results of active treatment trials, as well as the meta-analysis of control trials, we set the primary endpoint performance goal (PG $_6$ ) at 0.43.

Furthermore, the mean 6 month event rate from the meta-analysis of prior treatment studies is 0.38, with both the CHAMPION (0.37) and GUIDE-HF (0.31, NYHA class III) treatment groups with event rates lower than the mean. The lowest 6 month event rate across CardioMEMS control studies of 0.39 occurred in GUIDE-HF (NYHA class III), where modest use of SGLT2i occurred during the trial. We conservatively adjust this lowest observed control event rate down to 0.37 to account for increased SGLT2i utilization.

The table below outlines the data sources used to derive a PG for this endpoint.

Since patient level data was not available and summary data was limited in scope, analysis was based on the numbers of events reported from each study and the number of enrolled subjects was for the denominator, assuming all subjects were followed for the corresponding time period. Accordingly, the estimates are likely conservative underestimates of true rates since complete follow-up on all subjects was unlikely.

For studies reporting only 12-month rates, estimates of 6 month rates were estimated via an exponential distribution. For example, for a study with a reported enrollment n and 12-month rate,  $r_{12}$ , we calculated the 6 month rate,  $r_{6}$ , as:

$$r_6 = 1-\exp(\log_{10}(1-r_{12})/2)$$

where the division by two (2) accounts for a calculation of the rate for half the follow-up time. When possible, events of each type (HF related hospitalization and death) were calculated separately and summed to produce the composite event counts and the corresponding composite rate. Rates are calculated as numbers of events over numbers of subjects.

#### Active Treatment - updated 6 Month Rates with calculation details

| Study/Publication | Number of Subjects <sup>1</sup> | Events | Rate <sup>2</sup> | Details |
|---|---|---|---|---|
| CHAMPION [3] | 270 | 99 | 0.37 | - 6-month HFH rate reported as 0.31, yielding approx. 84 events - 15 deaths reported |

| | | | | - Adding calculated 6-month HFH events and deaths yields 99 events |
|---|---|---|---|---|
| MEMS PAS [4] | 1200 | 493 | 0.41 | - 6-month rate calculated via reported 12-month rate of 0.54 - Calculated 6-month HFH rate of 0.32, yielding 386 |
| | | | | events |
| | | | | - 107 deaths reported |
| | | | | - Adding calculated 6-month HFH events and deaths |
| | | | | yields 493 events |
| MEMS-HF [5] | 234 | 102 | 0.44 | - 6-month HFH calculated via reported 12-month rate of 0.60 |
| | | | | - Calculated 6-month HFH rate of 0.37, yielding 86 |
| | | | | events |
| | | | | - 16 deaths reported |
| | | | | - Adding calculated 6-month HFH and deaths yields<br>102 events |
| GUIDE-HF [6] – | 322 | 100 | 0.31 | - Reported 12 month rate of 0.431/0.089 for HFH/D, for composite of 0.52. |
| NYHA | | | | - Assuming exponential rate, calculated 6 month |
| class III only | | | | rate (events) is 0.31 (100) |
| , | | | | - Events calculated as 322 subjects x 0.31 |
| Estimate (CI) | | | | 0.38 (0.33, 0.44) |

<sup>1</sup> Numbers of subjects are those treated subjects estimated to be followed for 6-month events.

Altogether, for study success, the upper confidence bound of the observed event rate for the planned study must be less than the  $PG_6$  (0.43) and the observed event rate must be less than 0.37. Evaluating the upper bound of the confidence interval for the rate ensures that 1) the observed rate will be comparable to prior studies of active treatment (highest observed value = 0.44), 2) the observed rate will be less than the meta-analytic value derived from prior studies of treatment and control, and 3) the observed rate will be less than the lowest rate observed in the control studies (GUIDE HF). The added requirement for the observed event rate to be less than 0.37 provides further assurance that results are comparable to studies of prior CardioMEMS treatment.

The assumed PROACTIVE-HF population event rate is expected to be 0.34. This assumed event rate is lower than all prior active CardioMEMS treatment rates except for GUIDE-HF. While the contemporary GUIDE-HF study observed an event rate of 0.31 (NYHA Class III), PROACTIVE-HF has higher NTproBNP thresholds than the GUIDE-HF cohort and we expect subjects with higher NTproBNP levels to more closely align with subjects with a recent hospitalization, which have higher event rates. The mathematical statement of the null and alternative hypothesis is as follows:

 $Ho: r_6 \ge PG_6$ 

 $HA: r_6 < PG_6$ 

where  $r_6$  is the 6-month rate of primary endpoint events and  $PG_6$  is the performance goal. A value of 0.43 will be used for the goal. The null hypothesis will be rejected if the upper confidence bound for the rate is less than the performance goal, or equivalently, that the corresponding p-value from the hypothesis test is less than 0.025. An observed rate of less than 0.37 and rejection of the null hypothesis indicate that the observed rate is statistically less than the performance goal, indicating clinically acceptable results and

This document is confidential.


Controlled Document ID: 3903A.01, Effective Date 29-Oct-2018

<sup>&</sup>lt;sup>2</sup> Estimates for events are based on either reported results or are estimated from published figures. For studies reporting 12 month results, 6 month rates were estimated based on exponential rates.

study success. Analysis will be based on a Poisson regression approach for the number of events, with the log follow-up time as an offset term. Sensitivity analyses using a negative binomial approach to capture within-subject correlation will be performed.

The study will implant 450 subjects (combined in Cohort#2 and Cohort#3) leading to an expected evaluable cohort of 406 subjects. With a goal of 0.43 and a one-sided 0.025 alpha level, the study will have greater than 80% power assuming a population treatment rate of 0.34. Calculations are based on a one-sample Poisson rate test and were performed with PASS 2021.

#### 2.4.2. Additional Secondary Efficacy Endpoints

The first secondary efficacy endpoint is incidence of HF Hospitalizations or all-cause mortality at 12 months compared to a PG.

The mean 12 month event rate from the meta-analysis of prior control studies is 0.75, or 0.70 on an adjusted basis to account for SGLT-2i inclusion in the guidelines (Adjustment applied assuming 50% use of SGLT2i at the average hazard ratio observed across EMPEROR Preserved, EMPEROR REDUCED, DAPA-HF for NYHA III subjects.). A 12 month event rate of 0.70 represents a value just below the highest event rate observed across the CardioMEMS treatment studies (0.73 in MEMS-HF) and the upper bound of the overall meta-analytic treatment estimate (0.74). Taking the totality of results from the meta-analysis of active treatment trials, individual results of active treatment trials, as well as the meta-analysis of control trials, we set the secondary efficacy endpoint of performance goal (PG<sub>12</sub>) at 0.70.

Furthermore, the mean 12- month event rate from the meta-analysis of prior treatment studies is 0.64, with both the CHAMPION (0.6) and GUIDE-HF (0.52, NYHA class III) treatment groups with event rates lower than the mean. The lowest 12 month event rate across CardioMEMS control studies of 0.63 occurred in GUIDE-HF (NYHA class III only), where modest use of SGLT2i occurred during the trial. We conservatively adjust this lowest observed control event rate down to 0.59 to account for increased SGLT2i utilization.

The table below outlines the data sources used to derive a PG for this endpoint.

Active Treatment - updated 12 Month Rates with calculation details

| Study/Publication | Number of | Events | Rate <sup>2</sup> | Details |
|---|---|---|---|---|
| | Subjects <sup>1</sup> | | | |
| CHAMPION [7] | 270 | 162 | 0.60 | - HFH rate of 0.46, yielding approx. 124 events - Mortality rate of 0.14, yielding approx.38 events - Total events = 124 + 38 |
| MEMS PAS [4] | 1200 | 840 | 0.70 | - HFH rate of 0.54, yielding 648 events<br>- Mortality rate of 0.16, yielding 192 events<br>- Total events = 648 + 192 |
| MEMS-HF [5] | 234 | 171 | 0.73 | - HFH rate of 0.60, yielding 140 events<br>- Mortality rate of 0.13, yielding approx. 30 events<br>- Total events = 140 + 31 |
| GUIDE-HF [8] –<br>NYHA<br>class III only | 322 | 167 | 0.52 | - HFH rate of 0.431 + plus death rate of 0.0897<br>- Composite rate = 0.52<br>- Total events = 322 subjects x 0.52 |
| Estimate (CI) | | | | 0.64 (0.55, 0.74) |

Altogether, for study success, the upper confidence bound of the observed event rate for the planned study must be less than  $PG_{12}$  (0.70) and the observed event rate must be less than 0.59. Evaluating the upper

bound of the confidence interval for the rate ensures that 1) the observed rate will be comparable to prior studies of active treatment (highest observed value = 0.74), 2) the observed rate will be less than the meta-analytic value derived from prior studies of treatment and control, and 3) the observed rate will be less than the lowest rate observed in the control studies (GUIDE HF). The added requirement for the observed rate to be less than 0.59 provides further assurance that results are comparable to studies of prior treatment.

The assumed PROACTIVE-HF population event rate is expected to be 0.55. This assumed event rate is lower than all prior active CardioMEMS treatment rates except for GUIDE-HF. While the contemporary GUIDE-HF study (NYHA class III only) observed an event rate of 0.52, PROACTIVE-HF has higher NTproBNP thresholds than the GUIDE-HF cohort and we expect subjects with higher NTproBNP levels to more closely align with subjects with a recent hospitalization, which have higher event rates. The mathematical statement of the null and alternative hypothesis for the first secondary efficacy is as follows:

 $Ho: r_{12} \ge PG_{12}$  $Ha: r_{12} < PG_{12}$ 

where  $r_{12}$  is the 12 month rate of secondary endpoint events and  $PG_{12}$  is the performance goal. A value of 0.70 will be used for the goal. The null hypothesis will be rejected if the upper confidence bound for the rate is less than the performance goal, or equivalently, that the corresponding p-value from the hypothesis test is less than 0.025. An observed value of less than 0.59 and rejection of the null will indicate that the observed rate is statistically less than the performance goal, indicating clinically acceptable results. Analysis will be based on a Poisson regression approach for the number of events, with the log follow-up time as an offset term. Sensitivity analyses using a negative binomial approach to capture within-subject correlation will be performed.

Sample size calculations for the first secondary endpoint were performed in PASS 2021 and based on an assumed population event rate of 0.55, the sample size of 450 subjects would provide approximately 95% power for the secondary endpoint based on a one-sided 0.025 alpha level. If 406 subjects are followed for 12 months, approximately 95% power will be provided, so that the planned sample size is sufficient in light of potential attrition.

Formal hypothesis testing for the purposes of labeling claims for the first secondary efficacy endpoint will only be performed if the null hypothesis for the primary efficacy endpoint is successfully rejected.

This gatekeeping approach preserves the overall type I error rate. Any other calculated p-values and confidence intervals for secondary endpoints will be nominal, without adjustment for multiple comparisons.

#### 2.4.3. Primary Safety Endpoints

There are two primary safety endpoints.

Freedom from device or system related complications at 6 months will be tested against the null rate of 90%. A sample size of 450 patients provides greater than 95% power assuming a population rate of 95% for the freedom-from-event rates for device/system related complication at 6 months. Power would still be maintained at this level for an evaluable sample size of 406.

Similarly, Freedom from Pressure Sensor Failure at 6 months will be tested against the null rate of 95%. A sample size of 450 patients provides approximately greater than 95% power assuming a population rate of approximately 98.4%, for the pressure sensor failure at 6 months endpoint. Power would still be maintained at this level for an evaluable sample size of 406.

Mathematical statements of the null and alternative hypothesis for each test are as follows:

Ho: S1≥ PG<sub>s1</sub>

 $HA: S1 < PG_{s1}$ 

And

 $Ho: S2 \ge PG_{s2}$ 

*HA*: S2< PG<sub>s2</sub>

where S1 and S2 represent the freedom-from-event rates for device/system related complication at 6 months, and pressure sensor failure at 6 months respectively, and PGS1 and PGS2 represent the corresponding performance goals with values expressed as a proportion of 0.90 and 0.95 respectively.

Each of these will be assessed within among all patients who underwent a device implant by estimating freedom from the event of interest at 6 months by the Kaplan-Meier method. The proportion event free at 6 months and the corresponding two-sided 95% confidence interval will be compared to the null rate. We use a one-sample test of binomial proportions with a two-sided Type I error rate of 5% to estimate the power available for these analyses.

#### 2.5. Treatment Assignment & Blinding

This is an open-label study.

All subjects get implanted the Cordella PA Sensor in conjunction with a RHC procedure. The implantation takes place at the Implant Visit (V2). After deployment, the Sensor PAP is calibrated using a standard-of-care fluid-filled catheter for independent reference measurements. The calibration coefficients for that Sensor/Reader/Subject are stored in a database, allowing for accurate PAP calculations throughout the study duration.

Also, at the Implant Visit, eligible subjects will be provided with the commercially available Endotronix Cordella System to measure BP, HR, SpO2 and weight.

Subjects are observed until stable and discharged home with instructions their PAP measurements daily (same time each morning) along with their weight, BP, HR and SpO2, which are wirelessly transmitted to a secure website.

#### 2.6. Study Device

The investigational device is Cordella™ PA Sensor System.

The Cordella PA Sensor System comprises 7 subsystems that operate together to take daily PAP readings at a patient's home and transmit the results to a care provider for evaluation

- 1. Cordella Sensor
- 2. Cordella Delivery System
- 3. myCordella Patient Reader
- 4. Reader Dock
- 5. Cordella Calibration Equipment (CalEQ)
- 6. myCordella Tablet\*
- 7. Cordella Data Analysis Platform (CDAP)

For use in the proposed clinical trial, Endotronix intends to use the system in conjunction with Endotronix's commercial Cordella Heart Failure System (Cordella System). The Cordella System collects, records, and transmits physiologic data and communications from the patient at home to clinician(s) for assessment, patient communication, and patient-centered HF management.

It contains the following components:

- 1. myCordella Patient App
- 2. myCordella Patient Management Portal (PMP)
- 3. myCordella Tablet\*,\*\*
- 4. Up to 3 commercially available Medical Devices that patients use at home to collect data: weight, BP, HR and SpO2

The subjects are trained at the clinical site by a trained Clinical Site Delegate or Endotronix representatives on the set up and use of the Cordella System during the Screening/Enrollment Visit and for the the Cordella PA Sensor System at the Implant Visit (V2). Visits to the subject's home by an Endotronix Representative may be required throughout the study to provide troubleshooting, servicing, and maintenance of the system.

More detailed information about the study device can be found in Section 2 of the protocol.

#### 2.7. Study Procedures and Time and Event Schedule

For an overview of the timing of the clinical and laboratory measurements see Appendix 1: Time and Event Schedule.

<sup>\*</sup> the myCordella Tablet for the Cordella System and CorPASS systems are one and the same.

<sup>\*\*</sup> not a medical device in accordance with the 21st Century Cures Act.

## 3. Endpoints

#### 3.1. Primary Efficacy Endpoint

The primary efficacy endpoint is the 6 month incidence of HF related Hospitalizations (HFH) or all-cause mortalities.

#### 3.2. Primary Safety Endpoints

- 1. Freedom from device/system related complication at 6 months
- 2. Freedom from pressure sensor failure at 6 months

#### 3.3. Secondary Efficacy Endpoints

- 1. Incidence of HF Hospitalizations or all-cause mortality at 12 months
- 2. Number of HF Hospitalizations at 6 and 12 months post-implant compared to the number of HF Hospitalizations in the 6 and 12 months prior to implant
- 3. Comparison of the number of HF Hospitalizations or Emergency Department/ Hospital Outpatient V diuretic visits of Cohort #1 and Cohort #2 + #3 at 6 and 12 months post implant
- Change of N-terminal pro B-type Natriuretic Peptide (NT-proBNP) from Baseline through 6 and 12 months
- 5. Combined outcome of:
  - a. First and recurrent HF Hospitalizations
  - b. Heart failure Emergency Department/ Hospital Outpatient IV diuretic visits
  - c. all-cause mortality
- at 6 months, added together with equal weighting into a total number of events.
- 6. Heart failure hospitalization or HF Emergency Department / Hospital Outpatient IV diuretic visits at 6 and 12 month
- 7. Cardiac and all-cause mortality
- 8. Days Alive and Out of Hospital (DAOH)
- 9. Intravenous (IV) diuretic visits
- 10. Heart failure related Medication changes
- 11. Change in PAP:
  - a. From Baseline through 6 and 12 months in subjects with a baseline mPAP
    - i. above target range
    - ii. within or below target range
    - iii. Overall
  - b. Before and after 6-Minute Walk Test
- 12. Percentage of device success as documented by ability of the System to successfully transmit PAP data
- 13. Subject Outcome Measures, measured by Kansas City Cardiomyopathy Questionnaire (KCCQ)
- 14. Functional status improvement, as measured by NYHA and 6-Minute Walk Test
- 15. Health Economic Analysis (will be covered separately)

#### 3.4. **Secondary Safety Endpoints**

- 1. Pressure sensor failure rate throughout the study
- 2. Frequency of serious adverse events throughout the study
- 3. Frequency of implant procedure and procedure related adverse events and serious adverse events

### 4. Analysis Sets

#### 4.1. Enrolled Set

The Enrolled Set will include all subjects enrolled from Cohort #2 and #3. Screen failures are not part of this set. Subjects with either 'Did the Eligibility Committee approve the subject for Implant?' = 'No' (Form: 'Informed Consent') or 'Is subject eligible to participate in this study?' = 'No' (Form 'Eligibility') will be considered as screen failure. For rescreened patients, the previous patient number will be considered as screen failure, and the rescreened patient number will be included in enrolled set. Unless specified otherwise, this set will be used for subject listings and summaries of subject disposition.

#### 4.2. Intent-to-Treat Population

The Intent-to-Treat Population (ITT) will include all enrolled subjects intended to receive the Cordella PA Sensor who entered the Cath Lab, including those in whom Implant Procedure is not attempted for whatever reason (e.g. Cordella PA Sensor Implant cannot be performed due to anatomical reasons) from Cohort #2 and #3. Subjects in this population in whom the Cordella PA Sensor Implant is not attempted will be followed through 30 days for safety purposes. The ITT will be used for all analyses of safety endpoints. Efficacy analysis will not be performed on the ITT population.

#### 4.3. Modified Intent-to-Treat Population (mITT)

The Modified Intent-to-Treat Population (mITT) will include all implanted subjects from Cohort #2 and Cohort #3. All primary and secondary efficacy analyses as well as primary safety analyses will be performed on the mITT.

#### 4.4. Per Protocol Population

The Per Protocol Population (PP) will include all mITT subjects without any major protocol deviations. All primary and secondary safety and efficacy analyses will be performed in addition on PP population. If PP and mITT populations will be identical, analysis will be performed based on mITT only.

#### 4.5. Cohort #1 Population

This population will include all Cohort #1 (previously enrolled Control Arm) implanted subjects and will be reported separately for all applicable tables, figures and listings.

#### 4.6. Comparison Population

This population will include all implanted subjects from Cohort #1, Cohort #2 and #3. The Comparison Population will be used for analysis of secondary efficacy endpoint #3.

#### 4.7. Protocol Deviations

Sponsor will assess the protocol deviations as minor or major and provide this information to Syneos Health prior to date of cut-off, main analysis, and prior to database lock for the follow-up (final) analysis.

## 5. General Aspects for Statistical Analysis

#### 5.1. General Methods

- Unless otherwise specified, summaries will be presented by cohort (cohort #2 vs cohort #3) and overall
- Continuous variables will be summarized using the number of observations (n), mean, standard deviation (SD), median, minimum, and maximum. Categorical variables will be summarized using number of observations (n), frequency and percentages of subjects.
- All relevant subject data will be included in listings. All subjects entered into the database will be included in subject data listings, except screen failures. A separate listing will present the screen failures along with the inclusion criteria they failed and/or exclusion criteria they met. All listings except 16.2.3.x will be repeated for Cohort #1 population.
- In case of multiple assessments at a given time point (planned, repeat, unscheduled) the planned visit will be used for the analysis. For the definition of the baseline value, the last available value (e.g. unscheduled) prior to implant of Cordella PA Sensor will be used.

#### 5.2. Key Definitions

#### <u>Age</u>

Age at screening is derived in the database and this value will be used for all analyses.

#### <u>Definition of Baseline for safety assessments</u>

Baseline will be defined as the last available value prior to the implant of Cordella PA Sensor and may be at any visit between Screening (V1) and Cordella PA Sensor Implant Visit (V2).

#### Definition of Baseline for PAP measurements

Baseline will be defined as value at Implant Visit (V2) obtained before discharge.

## Change from Baseline

Absolute change from baseline:

Absolute change = Post-baseline value -baseline value

#### Time to Onset of AE

Time to onset of AE [days] = Date of start of AE - Date of implant of Cordella PA Sensor + 1

#### Start Day of concomitant medication

If medication starts before date of implant of Cordella PA Sensor:

Start Day of Medication = Date of start of medication – Date of implant of Cordella PA Sensor If medication starts at/after date of implant of Cordella PA Sensor

Start Day of Medication = Date of start of medication – Date of implant of Cordella PA Sensor + 1 Incomplete start dates of medication will not be imputed. Start day of medication will be missing.

#### Stop Day of concomitant medication

If medication stoped before date of implant of Cordella PA Sensor:

Stop Day of Medication = Date of end of medication – Date of implant of Cordella PA Sensor If medication stops at/after date of implant of Cordella PA Sensor

This document is confidential.


Controlled Document ID: 3903A.01, Effective Date 29-Oct-2018

Stop Day of Medication = Date of end of medication – Date of implant of Cordella PA Sensor + 1 Incomplete end dates of medication will not be imputed. Stop day of medication will be missing.

#### Definition of study completed/discontinued/ongoing

A subject will be defined as study 'completed' / discontinued' based on the eCRF information. At the time of the pre-defined main analysis, subjects which are ongoing at date of cut-off will be counted as 'ongoing'.

#### Time since first diagnosis of heart failure

Time since diagnosis [months] = ((Date of Screening – Date of first HF diagnosis)+1)/30

#### Exposure time:

which would be exact 6 or 12 months (180 or 365 days respective) post-implant visit for subjects who are still in the study at/after this timepoint.

which would be [date of last available date – date of Implant visit + 1] for subjects who withdraw from study prior to month 6 or 12 (180 or 365 days respective) post-implant visit.

#### 5.3. Missing Data

It is anticipated that there will be little or no missing data that would impact the ability to assess the primary endpoint. The primary efficacy analysis will be based on the mITT population and the primary safety analyses will be based on the population of subjects who underwent a device implant. The primary analysis methods naturally handle missing data by censoring subjects who have dropped out. For the primary safety analyses, the endpoints can be considered as dichotomous and the extreme cases as well as a tipping point analysis can be presented.

For all other analysis, missing data will not be replaced.

#### 5.4. Visit Windows

Every attempt should be made to perform evaluations at the designated time points. However, for visits conducted at Month 1 and 3 there is a window of +/-7 days, for visits at Month 6 there is a window of +/-14 days and after Month 6 (Month 12, 18, 24 and Year 3) there is a window of +/-30 days. All visits will be summarized according to the nominal visit.

#### 5.5. Pooling of Sites

Subjects will be pooled across sites for analysis of study endpoints. Sites with at least 20 subjects will retain their identities. Smaller sites will be ranked in decreasing order of size (site identification numbers, smallest first, will be used to break ties) and cumulatively pooled until pooled sites of no less than 10 subjects are achieved. After this pooling process, it will be tested for homogeneity in the treatment effects across site by using the same poisson model for primary endpoint but to add pooled site as a covariate. The homogeneity test will be conducted at the 0.15 level effect for pooled\_site.

run;

In case homogeneity in the rate across sites is not given, an explorative analysis will be performed as posthoc analysis, to evaluate in a first step what are the differences between the sites which may lead to different rates across sites. The possible factors will be evaluated during this exploratory analysis. In a second step a more complex analysis, e.g. Bayesian hierarchical model of HF event rates across pooled sites which is

This document is confidential.


Controlled Document ID: 3903A.01, Effective Date 29-Oct-2018

essentially treating site as a random effect could be performed. The final decision on the analysis to be performed will be evaluated outside of this SAP. Pooling of sites will be based on the mITT and PP populations.

#### 5.6. Subgroups

Subgroup analysis are planned to be performed by sex (female/male) and heart failure ejection fraction (HFrEF/HFpEF).

Heart failure ejection fraction will be defined based on the echocardiogram parameter: LVEF (%). If LVEF values are <= 40 then it is 'HFrEF', otherwise if LVEF values is >=50 then it is 'HFpEF'. A separate look will be at the LVEF values is > 40 - < 50 as a HFpEF subgroup.

Subgroup analysis is planned for efficacy and safety endpoints, subject disposition, demographics and other baseline characteristics, prior and concomitant medication.

### 6. Demographic, Other Baseline Characteristics and Medication

#### 6.1. Subject Disposition and Withdrawals

Subject disposition will be summarized by presenting the number and percentage of subjects eligible for the study, number of subjects in each analysis set, subjects completed the Month 6, V5 visit, subjects completed the Month 12, V6 visit, and completed or discontinued from the study together with the primary reason for premature termination, compliance with taking Cordella System daily reading per protocol. Additionally, presentation will be done by site.

Major protocol deviations will be summarized. In addition, a table will be generated summarizing the number of percentage of patients with a protocol deviation due to COVID-19.

Furthermore, the number of subjects excluded from each analysis set will be summarized by reason for exclusion.

Subject status at the study visits described in Appendix 1: Time and Event Schedule will be summarized presenting number of subjects alive, number of subjects with alive status (inpatient hospitalization/out subject), and number of subject with out status (home/rehabilitation centre/other) by visit.

In addition, subject training on Cordella system at implant visit will be presented in a separate table.

All data will be listed.

#### 6.2. Demographic

Demographic (age, gender, race, ethnicity, height, weight, and BMI), heart failure ejection fraction, and smoking history, will be presented in a summary table for mITT, ITT and PP population.

All data will be listed.

#### 6.3. Medical History and Concomitant Diseases

Medical history data will be summarized by category of medical condition for mITT, ITT and PP population. Medical history conditions with ongoing ticked 'No' will be considered as prior diseases, with ongoing ticked 'Yes' as concomitant diseases. In addition, all data will be listed.

Cardiac medical and surgical history data will be summarized by category of cardiac medical and surgical history for mITT, ITT and PP population. In addition, cardiac medical and surgical history will be listed.

#### 6.4. Other Baseline Characteristics

Summary table will be presented for 'Time since first diagnosis of heart failure', 'Type of first heart failure', 'Previous cardiovascular history', and 'Number of hospitalizations in past year for the cardiovascular reasons'

Cardiovascular history data will be summarized by category. In addition, cardiovascular history be listed.

#### 6.5. Medication

All medications will be coded using the WHO Drug Global B3, March 2019.

The number and percentage of subjects taking baseline and concomitant medications will be summarized overall by Anatomical Therapeutical Chemical (ATC) Levels 2 and 3 for mITT, ITT and PP population. All medication will be listed.

#### 6.5.1. Baseline Medication

Medications started prior to the date of implant will be summarized as 'Baseline' medications.

This document is confidential.


Controlled Document ID: 3903A.01, Effective Date 29-Oct-2018

#### 6.5.2. **Concomitant Medication**

Medications taken at/after the date of implant will be summarized as 'Concomitant' medications.

## 7. Efficacy

The population used for efficacy analyses will be the mITT. In addition, all efficacy analysis will be analyzed based on PP population and Cohort #1 population. For CEC related endpoints, tables and figures will be repeated using CEC adjudication results

#### 7.1. Primary Efficacy Endpoint and Analysis

The primary efficacy endpoint is the 6 month incidence of HF related hospitalizations (HFH) or all-cause mortality.

The information on mortality will be used as collected on the CRF, AE page with AE outcome = 'Death' or Study completion page with primary reason for discontinuation = 'Death'.

The information on HF hospitalizations will be used as collected on the CRF, Hospitalization page, only hospitalizations due to heart failure and stay at least 24 h will be considered as HF related hospitalizations

#### 7.1.1. Main analysis

The mathematical statement of the null and alternative hypothesis is as follows:

```
Ho: r_6 \ge PG_6
HA: r_6 < PG_6
```

will be used for the goal. The null hypothesis will be rejected if the upper confidence bound for the rate is less than the performance goal, or equivalently, that the corresponding p-value from the hypothesis test is less than 0.025. An observed rate of less than 0.37 and rejection of the null hypothesis indicate that the observed rate is statistically less than the performance goal, indicating clinically acceptable results and study success. Analysis will be based on a Poisson regression approach for the number of events, with the exposure time as an offset term, where  $r_6$  is the 6-month rate of primary endpoint events and  $PG_6$  is the performance goal. A value of 0.43 will be used for the goal.

The test will be based on each subject's total number of events, treatment arm, and exposure time, where a subject's exposure is the time to death, early study discontinuation or 6 months, whichever is smaller.

```
proc genmod data = xxx;
```

```
model number of events = dummy /*(dummy variable)*/ / noint type3 dist=poisson
offset=log(exposure_time);
run;
```

All events until day x, which would be exact 6 months (180 days) post-implant visit would be summarized by cohort. The estimated 6 month incidence of HF related hospitalizations (HFH) or all-cause mortality, along with the 2-sided 95% Cls for the estimated will be presented, and p-value from the hypothesis test. The presentation will also include number of HFH, all-cause mortality, total number of both events, and subjects' event rate of HFH or all-cause mortality is calculated as the total number of observed events per subject divided by the (subject's observed exposure time/180) from implant through 6 months, where a subject's exposure is the time to death, early study discontinuation or 6 months (180 days) post implant visit, whichever is the smallest.

#### 7.1.2. Sensitivity analysis

Sensitivity analyses using a negative binomial approach (with the same terms as the poisson model used in the main analysis) to capture within-subject correlation will be performed.

This document is confidential.


Controlled Document ID: 3903A.01, Effective Date 29-Oct-2018

#### 7.1.3. Supplementary analysis

Then main analysis will be repeated based on the PP population and Cohort #1 population. Interpretation of the p-values will be done in descriptive manner only.

In addition, HFH and all-cause mortality from CEC adjudication results will be analysed separately using same method as the main analysis in Section 7.1.1. Secondary Efficacy Endpoints and Analyses

7.1.4. Incidence of HF Hospitalizations or all-cause mortality at 12 months

The mathematical statement of the null and alternative hypothesis for the first secondary efficacy is as follows:

 $H_0: \mathbf{r}_{12} \ge PG_{12}$ 

 $H_A$ :  $r_{12} < PG_{12}$ 

where  $r_{12}$  is the 12 month rate of secondary endpoint events and  $PG_{12}$  is the performance goal. A value of 0.70 will be used for the goal. The null hypothesis will be rejected if the upper confidence bound for the rate is less than the performance goal, or equivalently, that the corresponding p-value from the hypothesis test is less than 0.025. An observed value of less than 0.59 and rejection of the null will indicate that the observed rate is statistically less than the performance goal, indicating clinically acceptable results.

Analysis will be based on a Poisson regression approach for the number of events, with the log follow-up time as an offset term. Sensitivity analyses using a negative binomial approach to capture within-subject correlation will be performed.

12 month incidence of HF related hospitalizations (HFH) or all-cause mortality will be analyzed on the mITT, PP and Cohort #1 population in a similar manner to the primary efficacy endpoint.

7.1.5. Number of HF Hospitalizations at 6 and 12 months post-implant compared to the number of HF Hospitalizations in the 6 and 12 months prior to implant

Heart Failure hospitalizations will be summarized by cohort presenting number of subjects without any hospitalizations at 6 and 12 months post-implant visit, number of subjects with any hospitalizations at 6 and 12 months post-implant visit, number of hospitalizations per subject at 6 and 12 months post-implant visit, and mean number of hospitalizations per subjects at 6 and 12 months post-implant visit. Similar presentation will be done based on the CRF information on the number of hospitalizations in the 6 and 12 months prior to implant. 95 % Clopper-Pearson confidence interval (CI) will be provided in addition for the frequencies as applicable. In additional, Wilcoxon rank sum tests will be performed to compare the number of hospitalizations per subject at 12 months post-implant visit with 12 months prior-implant visit, and compare the number of hospitalizations per subject at 6 months post-implant visit with 6 months prior-implant visit.

The 6 and 12 months timepoint is independently of visit information and is calculated as:

All events until day x, which would be exact 6 or 12 months (180 or 365 days respective) post-implant visit would be summarized.

All events happened between day x and implant visit, which is exact 6 or 12 months (-180 or -365 days respective) pre-implant visit. Analysis will be done based on mITT population, PP population, and Cohort #1 population. Prior to the date of cut-off for the main analysis, it will be confirmed, if analysis based on PP population will be required.

7.1.6. Comparison of the number of HF Hospitalizations or Emergency Department/ Hospital Outpatient IV diuretic visits of Cohort #1 and Cohort #2 + Cohort #3 at 6 and 12 month post implant

The rate of mortality and HF hospitalizations or HF emergency department/hospital outpatient IV diuretic visits in each cohort at 6 or 12 month is calculated as the total number of observed events in each cohort divided by the (total observed exposure time/180 or 365) in each cohort from implant visit through 6 months or 12 months.

The information on mortality will be used as collected on the CRF, AE page with AE outcome = 'Death' or Study completion page with primary reason for discontinuation = 'Death'. The information on HF hospitalizations will be used as collected on the CRF, Hospitalization page, emergency department/hospital outpatient IV diuretic visits will be used as collected on the CRF, AE page with AEs resulted in = 'Emergency Department (ED) visit'/ Hospitalization'/ 'Urgent, unscheduled outpatient office/practice' for AE categorized as 'Heart failure'.

The Cohort #1 and Cohort #2 + Cohort #3 subjects will then be compared with respect to rate of events per unit time using poisson regression. The test will be based on each subject's total number of events, treatment arm, and exposure time, where a subject's exposure is the time to death, early study discontinuation or 6 or 12 months, whichever is smaller.

Let  $\lambda_1$  be the rate of events per 6/12 moth on the Cohort #1 and let  $\lambda_2$  be the rate of events per 6/12 month on the Cohort #2 + Cohort #3. The null hypothesis is  $H_0$ :  $\lambda_1 \leq \lambda_2$  and the alternative hypothesis is  $H_1$ :  $\lambda_1 > \lambda_2$ .

The poisson regression calculation provides a one-sided p-value for the null hypothesis that the rate in the Cohort #1 is less than or equal to the rate in the Cohort #2 + Cohort #3.. The resulting p-values will be seen as explanatory.

proc genmod data = xxx;

class trt;

model number of events = trt/ type3 dist= poisson offset=log(exposure\_time);

run;

Analysis will be done based on the Comparison population.

7.1.7. Change of NT-proBNP from Baseline through 6 and 12 months

Change of NT-proBNP from baseline through 6 and 12 months will be presented by means of descriptive statistics at all study visits as described in Appendix 1: Time and Event Schedule.

Analysis will be done based on mITT population, PP population, and Cohort #1 population. Prior to the date of cut-off for the main analysis, it will be confirmed, if analysis based on PP population will be required.

7.1.8. Combined outcome of: a. First and recurrent HF Hospitalizations b. HF Emergency Department/ Hospital Outpatient IV diuretic visits c. all-cause mortality at 6 months

Number of total events will be calculated as the sum of the number of HF hospitalizations, HF emergency department/hospital outpatient IV diuretic visits and all-cause mortality. Both first and recurrent events will contribute to the total number. All events will be equal weighting.

This endpoint will be analyzed similarly as the primary endpoint in Section 7.1.1.

Analysis will be done based on mITT population, PP population and Cohort #1 population. Prior to the date of cut-off for the main analysis, it will be confirmed, if analysis based on PP population will be required.

# 7.1.9. Heart failure hospitalization or HF Emergency Department / Hospital Outpatient IV diuretic visits at 6 and 12 months

Number of total events will be calculated out of number of HF hospitalizations or HF emergency department/hospital outpatient IV diuretic visits at 6 and 12 months. First and recurrent events will account to the total number. All events will be equal weighting.

This endpoint will be analyzed similarly as the primary endpoint in Section 7.1.1.

In addition, time to first HF hospitalization/ time to first HF emergency department/hospital outpatient IV diuretic visit in days will be defined as the time from date of Implant visit to the date of the event. In case of no event during the observation period, subject will be censored on the last available date.

Definition of time to first HF hospitalization (days):

In case of event, time to first HF hospitalization = [(Date of event – date of Implant visit) + 1]

In case of no event, time to HF hospitalization = [(Date of last available date – date of Implant visit) + 1], this data will be censored.

Definition of time to first HF emergency department/hospital outpatient IV diuretic visit (days):

In case of event, time to first HF emergency department/hospital outpatient IV diuretic visit = [(Date of event – date of Implant visit) + 1]

In case of no event, time to HF emergency department/hospital outpatient IV diuretic visit = [(Date of last available date – date of Implant visit) + 1], this data will be censored.

Median duration of time to first HF hospitalization, time to first HF emergency department/hospital outpatient IV diuretic visit and respective 95% Cls will be reported using Kaplan Meier estimator and Kaplan Meier plot.

Time to HF hospitalization and time to HF emergency department/hospital outpatient IV diuretic visit will be listed.

Analysis will be done based on mITT population, PP population, and Cohort #1 population. Prior to the date of cut-off for the main analysis, it will be confirmed, if analysis based on PP population will be required.

#### 7.1.10. Cardiac and all-cause mortality

Time to all-cause mortality in days will be defined as the time from date of Implant visit to the date of the death. In case of no death during the observation period, subject will be censored on the last available date known alive.

Similarly, time to cardiac mortality in days will be defined as the time from date of Implant visit to the date of the cardiac death. In case of no cardiac death during the observation period, subject will be censored on the last available date known without cardiac death event.

Definition of time to death (days):

In case of event, time to death = [(Date of death – date of Implant visit) + 1]

In case of no event, time to death = [(Last available date – date of Implant visit) + 1], this data will be censored.

Definition of time to cardiac death (days):

This document is confidential.


Controlled Document ID: 3903A.01, Effective Date 29-Oct-2018

In case of event, time to cardiac death = [(Date of cardiac death – date of Implant visit) + 1]

In case of no event, time to cardiac death = [(Last available date without cardiac death event – date of Implant visit) + 1], this data will be censored.

Time to death/cardiac death will be listed and summarized by descriptive statistics.

Median duration of time to death and respective 95% Cls will be reported using Kaplan Meier estimator and Kaplan Meier plot.

Analysis will be done based on mITT population, PP population, and Cohort #1 population. Prior to the date of cut-off for the main analysis, it will be confirmed, if analysis based on PP population will be required.

#### 7.1.11. Days Alive and Out of Hospital (DAOH)

Days Alive and Out of Hospital (DAOH) calculated by subtracting days in hospital from total exposure time, where a subject's exposure is the time to death, early study discontinuation or 6 or 12 months, respectively, whichever is the smallest will be presented by means of descriptive statistics at 6 and 12 months post-implant visit.

Analysis will be done based on mITT population, PP population, and Cohort #1 population. Prior to the date of cut-off for the main analysis, it will be confirmed, if analysis based on PP population will be required.

#### 7.1.12. Hospital Outpatient IV diuretic visits

This endpoint will be analyzed similarly as the primary endpoint in Section 7.1.1.

Analysis will be done based on mITT population, PP population, and Cohort #1 population. Prior to the date of cut-off for the main analysis, it will be confirmed, if analysis based on PP population will be required.

#### 7.1.13. Heart failure related medication changes

Heart failure related medication change since last visit is collected via eCRF 'Has there been a change in the cardiovascular medication since last visit' and will be summarized by visit presenting the number and percentage of subjects with and without any change in HF medication.

Analysis will be done based on mITT population, PP population, and Cohort #1 population. Prior to the date of cut-off for the main analysis, it will be confirmed, if analysis based on PP population will be required.

### 7.1.14. Change in PA pressure

Change from baseline in PAP parameters collected via CorPASS: pulmonary artery pressure systolic, pulmonary artery pressure diastolic, pulmonary artery pressure mean and pulse will be presented by treatment group by means of descriptive statistics at before and after 6-minute walk test.

mPAP will be summarized by 'Above target range', 'Within or below target range', and 'Overall' for subjects with a baseline mPAP, at all study visits as described in Appendix 1: Time and Event Schedule including post implant measurement, and sitting vs. supine measurements. Shifts in mPAP from baseline over all post-baseline visits will be presented. Target range of mPAP is 5-20 mmHg. When there are more than one available results collected on same visit, please use the earliest one.

Analysis will be done based on mITT population, and PP population. Prior to the date of cut-off for the main analysis, it will be confirmed, if analysis based on PP population will be required.

This document is confidential.


Controlled Document ID: 3903A.01, Effective Date 29-Oct-2018
# 7.1.15. Percentage of device success as documented by ability of the System to successfully transmit PAP data

For the analysis of this endpoint, external data, provided by Endotronix, will be used. The provided data will include information if the missing PAP data are due to the System issues.

Following derived parameters will be presented:

- A) Total overall number of days of data collection, defined as the sum of all planned collection days (until end of study for final analysis or date of early discontinuation or date of cut-off or date of V6, Month 12 for the main analysis, whichever is smaller) of all subjects, excluding the days with missing data collection due to the subject's missing data transmission.
- B) Number of days with missing overall successful transmission of the collected data due to the System issues, defined as the sum of all unavailable days due to the System issues (until end of study for final analysis or date of early discontinuation or date of cut-off or date of V6, Month 12 date for the main analysis, whichever is smaller) of all subjects
- Overall device success rate of transmission (%), defined as A-B/A \* 100
- Per subject device success rate will be calculated similar to the rules above, based on per subject data only.

Per subject device success rate will be presented by means of descriptive statistics, overall device success rate as percentage, other parameters will be presented using counts.

Presentation will be done overall as all parameters are transmitted together.

Analysis will be done based on mITT population, PP population, and Cohort #1 population. Prior to the date of cut-off for the main analysis, it will be confirmed, if analysis based on PP population will be required.

## 7.1.16. Subject Outcome Measures, measured by Quality of Life KCCQ questionnaire

The Quality of Life KCCQ questionnaire is a measure of health-related quality of life. Data will be collected at the study visits described in Appendix 1: Time and Event Schedule. For the analysis of this endpoint, external data, provided by Endotronix, will be used.

The KCCQ is a 23-item, refer to Protocol, section 14.4, self-administered instrument that quantifies physical function, symptoms (frequency, severity, and recent change), social function, self-efficacy and knowledge, and quality of life related to HF.

Out of 23-items, 10 scores will be calculated according to the rules in Appendix 2: The Kansas City Cardiomyopathy Questionnaire Scoring Instructions: Physical Limitation, Symptom Stability, Symptom Frequency, Symptom Burden, Total Symptom Score, Self-Efficacy, Quality of Life, Social Limitation, Overall Summary Score, Clinical Summary Score.

Presentation will be done by means of descriptive statistics including the absolute value and change from baseline by visit.

Analysis will be done based on mITT population, PP population, and Cohort #1 population. Prior to the date of cut-off for the main analysis, it will be confirmed, if analysis based on PP population will be required.

## 7.1.17. Functional status improvement measured by NYHA and 6-Minute Walk Test

NYHA functional classification: The subject's functional status is assessed by a qualified individual at the institution, who is not directly involved with this clinical trial, by utilizing the NYHA functional classification, described in the Protocol Appendix 14.2.

The NYHA functional classification categorizes the extent of heart failure by placing subjects in one of four (I, II, IV) categories based on how much they are limited during physical activity and symptoms of shortness of breath and/or angina.

This document is confidential.


Controlled Document ID: 3903A.01, Effective Date 29-Oct-2018

NYHA functional classification will be obtained at all study visits as described in Appendix 1: Time and Event Schedule and must be NYHA Class III for study entry.

Shifts in NYHA functional classification from baseline over all post-baseline visits will be presented.

Six (6) Minute Walk: Subjects complete a six (6) minute walk test at the study visits described in Appendix 1: Time and Event Schedule. Total distance walked (meters) will be collected and analyzed by means of descriptive statistics including the absolute value and change from baseline by visit.

Analysis will be done based on mITT population, PP population, and Cohort #1 population. Prior to the date of cut-off for the main analysis, it will be confirmed, if analysis based on PP population will be required.

## 8. Safety

The population used for safety analyses will be the ITT. Safety will be assessed on the basis of adverse events (AEs), clinical laboratory data, ECG parameters, Echocardiograms, physical examinations, and vital signs. Primary safety endpoint will be analyzed based on mITT. In addition, AEs will be analyzed based on Cohort #1 population. Primary safety endpoints will also be repeated on ITT, PP population and Cohort #1 population. Secondary safety endpoints will also be analyzed based on PP population and Cohort #1 population. For CEC related endpoints, tables and figures will be repeated using CEC adjudication results

Adverse events and other safety analyses will also be assessed. No formal statistical hypothesis tests will be conducted. Analyses will involve Kaplan-Meier curves for time to event outcomes, descriptive statistics (n, mean, standard deviation, median, minimum, and maximum) for quantitative outcomes, and count and frequency results for categorical outcomes.

Safety analysis will be performed in first line to address the safety endpoints:

## 8.1. Primary safety endpoint

## 8.1.1. Main analysis

There are two primary safety endpoints:

- 1) Freedom from device/system related complication at 6 months. Freedom from device or system related complications at 6 months will be tested against the null rate of 90%. The endpoint will be assessed based on the AE CRF page with adverse event type = 'Device / System-Related Complication'
- 2) Freedom from pressure sensor failure at 6 months. Freedom from Pressure Sensor Failure at 6 months will be tested against the null rate of 95%. The endpoint will be assessed based on the AE CRF page with adverse event type = 'Pressure Sensor Failure'

Each of these will be assessed within among all subjects who underwent a device implant by estimating freedom from the event of interest at 6 months by the Kaplan-Meier method.

Definition of time to event (days):

In case of event, time to event = [(Date of event - date of Implant visit) + 1]

In case of no event, time to event = [(Date of last available date or date of day 180 [6 months] – date of Implant visit) + 1], this data will be censored.

The event free rate and respective 95% Cis based on KM method will be compared to the null rate.

#### For endpoint 1:

H0: rate of freedom from device/system related complication at 6 months <= 90 %

H1: rate of freedom from device/system related complication at 6 months > 90

## For endpoint 2:

H0: rate of freedom from pressure sensor failure at 6 months <= 95 %

H1: rate of freedom from pressure sensor failure at 6 months > 95 %

#### 8.1.2. Sensitivity analysis

Two kinds of sensitivity analysis are planned to be performed for the imputation of missing values for the primary safety endpoints. Sensitivity analysis will be performed if the main analysis results show significant effect.

#### Extreme cases analysis:

In case a subject withdraws from study prior to 6 months follow-up visit and without experiencing previously 'device/system related complication' or 'pressure sensor failure' respectively, the subject will be defined as

This document is confidential.


Controlled Document ID: 3903A.01, Effective Date 29-Oct-2018

having experienced such an event for the 6 months analysis. Setting all missing events to 'Y' would be the only possible extreme cases value. After imputation, below analysis will be performed.

```
For endpoint 1:

proc freq data= xxx

tables freedom (Y/N) / binomial(exact p=0.90 level = 1);

run;

define level = 1 'no event = no device/system related complication'

For endpoint 2:

proc freq data= xxx

tables freedom (Y/N) / binomial(exact p=0.95 level = 1);

run;

define level = 1 'no event = no pressure sensor failure at 6 months'

Tipping point analysis:
```

If the null hypothesis is rejected for primary safety end point, a tipping point analysis will be conducted based on the binary response of freedom from event/with event at 6 months using similar manner as extreme cases analysis. For subjects withdraws from study prior to 6 months follow-up visit and without experiencing previously 'device/system related complication' or 'pressure sensor failure' respectively, setting all missing events to 'N', then gradually increasing the number of subjects with event at 6 months until null hypothesis is not rejected.

## 8.2. Secondary safety endpoints

- 1) Pressure sensor failure rate throughout the study
- 2) Frequency of serious adverse events throughout the study
- 3) Frequency of implant procedure and procedure related adverse events and serious adverse events

Both secondary endpoints will be evaluated based on the AEs information and covered by AEs outputs.

#### 8.3. Adverse Events

All collected adverse events (AEs) will be coded using MedDRA, version 24.0, to give a preferred term and a SOC term for each event and used for the analysis.

#### 8.3.1.1. Device deficiency (DD)

Device deficiency is collected on a separate eCRF page called 'Device deficiency'. Summary will include the number and percent of subjects experienced device deficiency, number and percent of subjects with device deficiency resulted in AE, and number and percent of subjects with potential unanticipated adverse device effect (UADE) due to device deficiency.

#### 8.3.2. Relationship

An AE is considered related, if the relationship to study procedure is documented as 'possibly related', or 'related'.

An AE is considered device/system related complication (DSRC), if the relationship to study device is documented as 'possible related' or 'related'.

An AE is considered related to implant procedure, if the relationship to implant procedure is documented as 'possibly related' or 'related'.

Missing and/or unknown relationship will be presented as separate category, if available.

This document is confidential.


Controlled Document ID: 3903A.01, Effective Date 29-Oct-2018

#### 8.3.3. Predefined AE categories

Following AE categories are predefined in the study protocol, refer to Section 14.6 of the protocol for more information:

- 1. ACUTE KIDNEY INJURY graded as Stage 1, Stage 2 and Stage 3b
- 2. BLEEDING graded as Life-threatening or disabling bleeding (BARC type 5 or BARC type 3b and 3c or BARC type 3b), Major bleeding (BARC type 3a), Minor bleeding (BARC type 2 or 3a, depending on the severity)
- CONDUCTION DISTURBANCES AND ARRHYTHMIAS
- 4. DEATH classified as Cardiovascular (CV) death, Non-cardiovascular death or undetermined cause of death.
- DEVICE / SYSTEM-RELATED COMPLICATION
- 6. HEART FAILURE (HF)
- 7. HEMOPTYSIS
- 8. MYOCARDIAL INFARCTION (MI) classified as Peri-procedural MI (≤72 h after the index procedure) or Spontaneous MI (>72 h after the index procedure)
- PRESSURE SENSOR FAILURE
- 10. PULMONARY EMBOLISM
- 11. PULMONARY OCCLUSION
- 12. RENAL DYSFUNCTION classified as Acute renal dysfunction or Chronic renal dysfunction
- 13. STROKE (Non-Fatal) AND TRANS ISCHEMIC ATTACK (TIA) classified as Stroke or TIA STROKE CLASSIFICATION as Ischemic, Hemorrhagic or undetermined STROKE DEFINITION as Disabling stroke or Non-disabling stroke
- 14. VASCULAR ACCESS SITE AND ACCESS-RELATED COMPLICATIONS classified as Major vascular complications or Minor vascular complications
- 15. VESSEL TRAUMA classified as Blunt injury or Penetrating injury
- 16. OTHER <specify>

All SAEs and some selected AEs will be sent for adjudication.

#### 8.3.4. Presentation

Tables will be presented as listed below.

- An overall summary of the number and percentage of subjects reporting AEs, serious AEs, study
  procedure related AEs, serious study procedure related AEs, AEs leading to withdrawal and AEs
  leading to death, DSRC, Unanticipated Adverse Device Effect (UADE), implant procedure related
  AEs, serious implant procedure related AEs, and subjects who died.
- Predefined AEs by category
- AEs, overall and by SOC and preferred term
- Serious AEs, overall and by SOC and preferred term
- Serious AEs, overall and by preferred term
- Serious AEs by Seriousness Criteria
- Serious predefined AEs by category

This document is confidential.


Controlled Document ID: 3903A.01, Effective Date 29-Oct-2018

Statistical Analysis Plan for Interventional Studies Sponsor: Endotronix, Protocol No.: ETX-HFS-PA-03

• Study procedure related AEs, overall and by SOC and preferred term

Serious study procedure related AEs, overall and by SOC and preferred term

Implant procedure related AEs, overall and by SOC and preferred term

Serious implant procedure related AEs, overall and by SOC and preferred term

Study procedure related AEs by procedure type

AEs by maximum severity, overall and by SOC and preferred term

AEs by maximum relationship to implant procedure, overall and by SOC and preferred term

DSRC, overall and by SOC and preferred term

DSRC by maximum severity, overall and by SOC and preferred term

DSRC, by devices

UADE, overall and by SOC and preferred term

UADE by maximum severity, overall and by SOC and preferred term

UADE, by devices

• Implant procedure related AEs, overall and by SOC and preferred term

• Predefined AEs by relationships to device and study procedure from CEC adjudication results

AEs leading to study withdrawal, overall and by SOC and preferred term

Device deficiency will be presented as described in Section 8.3.1.1

 AEs, overall and by SOC and preferred term will be done for subjects with predefined AE category 'Pressure Sensor Failure'.

anticipated AEs, overall and by SOC and preferred term

anticipated AEs by maximum severity, overall and by SOC and preferred term

anticipated AEs by maximum relationship to implant procedure, overall and by SOC and preferred

term

unanticipated AEs, overall and by SOC and preferred term

unanticipated AEs by maximum severity, overall and by SOC and preferred term

- unanticipated AEs by maximum relationship to implant procedure, overall and by SOC and preferred term
- Other serious adverse events (AE) CEC adjudicated by system organ class and preferred term

Listings will be provided for all AEs, UADEs, DSRC, SAEs, anticipated AEs, unanticipated AEs, deaths, AEs leading to study withdrawal and predefined AEs by category. All collected data will be presented as available.

## 8.4. Laboratory Evaluations

All laboratory analyses will be performed by the local laboratory using standard assay methods. Laboratory evaluation is assessed at the study visits described in Appendix 1: Time and Event Schedule and includes chemistry, hematology, coagulation, Serum NT-pro BNP, and urinalysis with the following parameters:

## Chemistry

- Sodium
- Potassium
- Creatinine
- Total bilirubin
- Blood urea nitrogen (BUN)
- Urea
- Total protein
- Albumin
- CRP
- Aspartate aminotransferase (SGOT/AST)
- Alanine aminotransferase (SGPT/ALT)
- Cholesterol
- Uric acid

## Hematology

- Hemoglobin
- Hematocrit
- Leukocytes
- Platelets
- Lymphocytes

#### Coagulation

- INR (if indicated)
- aPTT

## NT-pro BNP

NT-pro BNP

#### **Urinalysis**

- pH
- Protein
- Glucose
- Ketones
- Occult blood
- RBC
- WBC
- Urobilinogen

This document is confidential.

- Bilirubin
- Specific gravity
  - Nitrite

## **Pregnancy test**

Urine pregnancy test

All laboratory results, including abnormal ranges, will be converted to the International System (SI) units, where applicable.

Summary tables consisting of normal, abnormal clinically significant (CS) and abnormal not clinically significant (NCS) for each parameter, by visit, will be provided. If a parameter has a missing value the result will be included in the summary table as missing.

All data will be included in data listings.

Pregnancy test data will be listed only.

## 8.5. Vital Signs

Vital signs (systolic blood pressure, diastolic blood pressure, heart rate, arterial oxygen saturation level (%), weight and BMI) are assessed at all study visits as described in Appendix 1: Time and Event Schedule. For vital signs parameters, absolute values and change from baseline will be presented by means of descriptive statistics at all scheduled study visits.

All data will be included in data listings.

## 8.6. Electrocardiogram (ECG)

A 12-lead electrocardiogram (ECG) (PR, RR, QRS, uncorrected QT, corrected QTcB, corrected QTcF) is assessed at the study visits described in Appendix 1: Time and Event Schedule. At each scheduled visit Investigator will provide overall ECG evaluation classifying the ECG as normal, abnormal NCS and abnormal CS.

Overall ECG evaluation by visit and shifts from baseline over all post-baseline results will be presented for overall ECG evaluation displaying normal, abnormal NCS and abnormal CS values.

All data will be included in data listings.

## 8.7. Echocardiogram

Echocardiogram is assessed at the study visits described in Appendix 1: Time and Event Schedule.

Following parameters will be evaluated:

- Left Ventricular Ejection Fraction (%) (LVEF)
- Left ventricular mass
- Left ventricular volume
- Left Ventricular End Diastolic Dimension (LVEDD)
- Left atrial size
- Left atrial volume
- Mitral regurgitation
- Systolic pulmonary artery pressure (sPAP)
- Diastolic pulmonary artery pressure (dPAP)
- Mean pulmonary artery pressure (mPAP)
- Tricuspid regurgitation Peak Velocity
- End Diastolic Pulmonary Regurgitation Gradients

This document is confidential.


Controlled Document ID: 3903A.01, Effective Date 29-Oct-2018

- Right atrial pressure (RAP)
- Overall Interpretation

At each visit Investigator will provide Overall interpretation evaluation classifying the Echocardiogram as normal, abnormal NCS and abnormal CS.

Overall interpretation by visit and shifts from screening to Visit 6 (Month 12) will be presented for overall interpretation displaying normal, abnormal NCS and abnormal CS values.

All data will be included in data listings.

## 8.8. Physical Examination

Complete physical examinations including body systems: general appearance, dermatological, lymphatic, head/ears/eyes/nose/throat (HEENT), chest/lungs, cardiovascular, abdomen, genitourinary/reproductive, musculoskeletal/extremities, neurologic/psychiatric and other) will be conducted at screening visits, Abbreviated physical examination will be conducted at all study visits as described in Appendix 1: Time and Event Schedule, collecting only the changes from screening assessment.

In addition, chest circumference will be collected at screening.

Physical examination data will be summarized at screening visit, all data will be listed only.

#### 9. **Interim Analyses**

Interim analysis is not planned.

## 10. Changes from Analysis Planned in Protocol

During the preparation of the SAP, it was realized that some additional analysis outside the protocol is needed. The respective analysis were introduced in the respective sections and are summarized below.

- 1) It was clarified that cardiac and all-cause mortality will be analyzed at 6 and 12 months post-implant visit, to be consistent with other efficacy analyses.
- 2) Two enrollment stopping rules will be considered during the study, both rules will be applied independently of each other and as well independent of the treatment group, see section 2.2. The enrollment stopping rules will ensure enrollment of sufficient number of subjects of certain population: at least 30 % women and at least 45 % HFpEF. This approach was previously confirmed by Sponsor with FDA.
- 3) Subgroup analysis was not clearly defined in the protocol: two population groups are of interest and were introduced in Section 5.6. This analysis is in line with the introduction of the enrollment stopping rules for the same populations, see Section 2.2.

## 11. Reference List

- 1. DSMB Statistical Analysis Plan Version 3.1 dated 07-Feb-2022
- 2. DSMB charter Version 4.0 dated 04-Mar-2022
- 3. Abraham, W. T., Adamson, P. B., Bourge, R. C., Aaron, M. F., Costanzo, M. R., Stevenson, L. W., CHAMPION Trial Study Group. (2011). Wireless pulmonary artery haemodynamic monitoring in chronic heart failure: a randomized controlled trial. Lancet, 377, 658-666.
- 4. Shavelle D. et al. Lower Rates of Heart Failure and All-Cause Hospitalizations During Pulmonary Artery Pressure-Guided Therapy for Ambulatory Heart Failure. Circ Heart Fail. 2020;13:e006863.
- 5. Angermann, C., Assmus, B., Anker, S.D., Asselbergs, F.W. Pulmonary artery pressureguided therapy in ambulatory patients with symptomatic heart failure: the CardioMEMS European Monitoring Study for Heart Failure (MEMS-HF). Eur J Heart Fail. 2020; 22 (10): 1891-1901
- 6. PMA P100045/S056B: FDA Summary of Safety and Effectiveness Data (SSED) CardioMEMS™ HF System
- 7. Lindenfeld, J.A., Zile, M, Desai, A.S., Bhatt, K, Adamson, P. B. Haemodynamic-guided management of heart failure (GUIDE-HF): a randomised controlled trial. Lancet, 2021; 398; 10304: 991-1001
- 8. PMA P100045 IDE G060187 December 2011 presentation to FDA Circulatory System Devices Advisory Panel. Slide 93-95

## 12. Programming Considerations

All tables, figures, listings (TFLs), and statistical analyses will be generated using SAS for Windows, Release 9.4 or higher (SAS Institute Inc., Cary, NC, USA). Computer-generated table, listing and figure output will adhere to the following specifications.

#### 12.1. General Considerations

- One SAS program will be created for each output.
- Each output will be stored in a separate file.
- Output files will be delivered in Word format (RTF). One portable document format pdf will be delivered for tables, listings, and figures.
- Numbering of TFLs will follow ICH E3 guidance

## 12.2. Table, Listing, and Figure Format

#### 12.2.1. General

- All TFLs will be produced in landscape A4 format, unless otherwise specified.
- All TFLs will be produced using the Courier New font, size 9 which is the smallest acceptable point size for the Regulatory Authorities.
- The data displays for all TFLs will have a minimum blank 1-inch margin on all 4 sides.
- Headers and footers for figures will be in Courier New font, size 8 which is the smallest acceptable point size for the Regulatory Authorities.
- Legends will be used for all figures with more than 1 variable, group, or item displayed.
- TFLs will be in black and white (no color), unless otherwise specified
- Specialized text styles, such as bolding, italics, borders, shading, and superscripted and subscripted text, will not be used in the TFLs, unless otherwise specified. On some occasions, superscripts 1, 2, or 3 may be used.
- Only standard keyboard characters will be used in the TFLs. Special characters, such as non-printable control characters, printer-specific, or font-specific characters, will not be used.
  Hexadecimal-derived characters will be used, where possible, if they are appropriate to help display math symbols (e.g., µ).
- Mixed case will be used for all titles, footnotes, column headers, and programmer-supplied formats, as appropriate.

## 12.2.2. Headers

- All output should have the following header at the top left of each page:
- Endotronix Protocol ETX-HFS-PA-03 (Syneos Health study number 7000235)

This document is confidential.

- Draft/Final/Follow-up Run
- All output should have Pagen of Nat the top right corner of each page. TFLs are internally paginated in relation to the total length (i.e., the page number should appear sequentially as page n of N, where N is the total number of pages in the table).
- The date output was generated should appear along with the program name as a footer on each page.

## 12.2.3. Display Titles

Each output is identified by the designation and a numeral (i.e., Table 14.1.1). ICH E3 numbering
will be applied. The title is centered. The analysis set is identified on the line immediately following
the title.

First Line of Title
Second Line of Title if Needed
(ITT Analysis Set)

## 12.2.4. Body of the Data Display

#### 12.2.4.1. General Conventions

Data in columns of a table or listing are formatted as follows:

- Alphanumeric values are left-justified;
- Whole numbers (e.g., counts) are right-justified; and
- Numbers containing fractional portions are decimal aligned.

#### 12.2.4.2. Table Conventions

- Units will be included where available
- Unless otherwise specified, only those categories for which there is at least 1 subject represented in 1 or more groups are included.
- Where percentages are presented in these tables, zero percentages will not be presented and so counts of 0 will be presented as 0 and not as 0 (0%).
- A Missing category is added to each parameter for which information is not available for 1 or more subjects.
- Unless otherwise specified, the estimated mean and median for a set of values are printed out to 1
  more significant digit than the original values, and standard deviations are printed out to 2 more
  significant digits than the original values. The minimum and maximum should report the same
  significant digits as the original values.
- Percentage values are printed to one decimal place, in parentheses with no spaces, one space after the count (e.g., 7 (12.8%), 13 (5.4%)). Values that round down to 0.0 will be displayed as '<0.1'.</li>
   Unless otherwise noted, for all percentages, the number of subjects in the analysis set for the given

This document is confidential.

group who have an observation will be the denominator. Percentages after zero counts should not be displayed and percentages equating to 100% are presented as 100%, without decimal places.

• Where a category with a subheading (such as system organ class) has to be split over more than one page, output the subheading followed by "(cont)" at the top of each subsequent page. The overall summary statistics for the subheading should only be output on the first relevant page.

## 12.2.4.3. Listing Conventions

- Listings will be sorted for presentation by subject number, visit/collection day, and visit/collection time.
- Dates are printed in SAS DATE9.format ("ddMMMyyyy": 01JUL2000). Missing portions of dates are represented on subject listings as dashes (--JUL2000).
- All observed time values are to be presented using a 24-hour clock HH:MM or HH:MM:SS format (e.g., 11:26:45, or 11:26). Time will only be reported if it was measured as part of the study.
- Units will be included where available

## 12.2.5. Footnotes

- A solid line spanning the margins will separate the body of the data display from the footnotes.
- All footnotes will be left justified with single-line spacing immediately below the solid line underneath the data display.
- Subject specific footnotes are avoided, where possible.
- Footnotes will be used sparingly and add value to the table, figure, or listing. If more than six lines of footnotes are planned, then a cover page will be used to display footnotes.
- The last line of the footnote section will be a standard source line that indicates the name of the program used to produce the data display, date the program was run, and the listing source (i.e., 'Program: myprogram.sas Listing source: 16.x.y.z').

## 13. Quality Control

SAS programs are developed to produce output such as analysis data sets, summary tables, data listings, figures or statistical analyses.

Syneos Health SOPs Developing Statistical Programming Specifications (3906), Developing Statistical Programs (3907) and Conducting the Transfer of Biostatistical Deliverables (3908) describe the quality control procedures that are performed for all SAS programs and output. Quality control is defined here as the operational techniques and activities undertaken to verify that the SAS programs produce the output by checking for their logic, efficiency and commenting and by review of the produced output.

## 14. Index of Tables

| Table | | |
|---|---|---|
| Number | Name | Analysis Set |
| | | , |
| | Demographic Data Summary Tables | |
| 14.1.1.1 | | Enrolled Population |
| | | Cohort #1 |
| | | Population |
| 14.1.1.2 | Subject disposition by site and pooled sites | Enrolled Population |
| | | Cohort #1 |
| | | Population |
| 14.1.1.3 | Subject status | mITT Population |
| 14.1.1.3.1 | | Cohort #1 |
| | , | population |
| 14.1.1.4 | Subject training pre-implant | mITT Population |
| 14.1.1.4.1 | | Cohort #1 |
| | | Population |
| | Protocol Deviations | |
| 14.1.2.1 | | Enrolled Population |
| | | Enrolled Population |
| | | Enrolled Population |
| | | • |
| 14.1.3.1.1 | | mITT Population |
| | | ITT Population |
| 14.1.3.1.3 | Subject demographic and baseline characteristics, | mITT Population |
| 14.1.3.1.4 | | mITT Population |
| | | ' |
| 14.1.3.1.5 | | Per Protocol |
| | | Population |
| 14.1.3.1.6 | Subject demographic and baseline characteristics | Cohort #1<br>Population |
| | Other Baseline Disease Characteristics | · · · · |
| 14 1 3 2 1 | | mITT Population |
| | Cardiovascular history - overall summary | ITT Population |
| | | mITT Population |
| 11.1.0.2.0 | | IIII Opalation |
| 14 1 3 2 4 | | mITT Population |
| | | min i opalation |
| 14.1.3.2.5 | | Per Protocol |
| | | Population |
| 14.1.3.2.6 | Cardiovascular history - overall summary | Cohort #1 |
| | , | Population |
| 14.1.3.2.7 | Cardiovascular history | mITT Population |
| | | ITT Population |
| | | mITT Population |
| 14.1.3.2.10 | Cardiovascular history, stratified by heart failure | mITT Population |
| 14.1.3.2.11 | | Per Protocol |
| | | Population |
| | 14.1.1.1<br>14.1.1.1<br>14.1.1.2<br>14.1.1.2.1<br>14.1.1.3<br>14.1.1.4<br>14.1.1.4.1<br>14.1.1.4.1<br>14.1.2.1<br>14.1.2.2<br>14.1.2.3<br>14.1.3.1.1<br>14.1.3.1.2<br>14.1.3.1.3<br>14.1.3.1.6<br>14.1.3.2.1<br>14.1.3.2.1<br>14.1.3.2.1<br>14.1.3.2.2<br>14.1.3.2.3<br>14.1.3.2.3<br>14.1.3.2.3 | Demographic Data Summary Tables |

This document is confidential.

SAP Version: 3.0 dated 17-Aug-2023 Controlled Document ID: **3903A.01**, Effective Date 29-Oct-2018

| | Table | | |
|---|---|---|---|
| Header | Number | Name | Analysis Set |
| | 14.1.3.2.12 | Cardiovascular history | Cohort #1 |
| | | ,,, , | Population |
| 14.1.3.3 | | Medical History | <b>'</b> |
| | 14.1.3.3.1 | Medical history | mITT Population |
| | 14.1.3.3.2 | Medical history | ITT Population |
| | 14.1.3.3.3 | Medical history | Per Protocol |
| | | , , | Population |
| | 14.1.3.3.4 | Medical history | Cohort #1 |
| | | | Population |
| | 14.1.3.3.5 | Cardiac/medical and surgical history | mITT Population |
| | 14.1.3.3.6 | Cardiac/medical and surgical history | ITT Population |
| | 14.1.3.3.7 | Cardiac/medical and surgical history | Per Protocol |
| | | | Population |
| | 14.1.3.3.8 | Cardiac/medical and surgical history | Cohort #1 |
| | | j , | Population |
| 14.1.4 | | Medications | , |
| | 14.1.4.1 | Baseline medications | mITT Population |
| | 14.1.4.2 | Baseline medications | ITT Population |
| | 14.1.4.3 | Baseline medications, stratified by sex | mITT Population |
| | 14.1.4.4 | Baseline medications, stratified by heart failure | mITT Population |
| | | ejection fraction | ' |
| | 14.1.4.5 | Baseline medications | Per Protocol |
| | | | Population |
| | 14.1.4.6 | Baseline medications | Cohort #1 |
| | | | Population |
| | 14.1.4.7 | Concomitant medications | mITT Population |
| | 14.1.4.8 | Concomitant medications | ITT Population |
| | 14.1.4.9 | Concomitant medications, stratified by sex | mITT Population |
| | 14.1.4.10 | Concomitant medications, stratified by heart failure | mITT Population |
| | | ejection fraction | · |
| | 14.1.4.11 | Concomitant medications | Per Protocol |
| | | | Population |
| | 14.1.4.12 | Concomitant medications | Cohort #1 |
| | | | Population |
| | 14.1.4.13 | Concomitant medication by category | mITT Population |
| | 14.1.4.14 | Concomitant medication by category | Cohort #1 |
| 110 | | | Population |
| 14.2 | | Efficacy Data Summary Figures and Tables | |
| 14.2.1 | 1440444 | Primary Efficacy Parameter | |
| | 14.2.1.1.1 | 6-month incidence of HF hospitalizations (HFH) or | mITT Population |
| | 440444 | all-cause mortalities | ITT D ! !! |
| | 14.2.1.1.1a | SAS-Output: 6-month incidence of HF | mITT Population |
| | 140110 | hospitalizations (HFH) or all-cause mortalities | mITT Danislatias |
| | 14.2.1.1.2 | 6-month incidence of HF hospitalizations (HFH) or | mITT Population |
| <u> </u> | 14.2.1.1.2a | all-cause mortalities, stratified by sex SAS-Output: 6-month incidence of HF | mITT Danulation |
| 1 | 14.2.1.1.2a | | mITT Population |
| | | hospitalizations (HFH) or all-cause mortalities, | |
| | 14.2.1.1.3 | stratified by sex 6-month incidence of HF hospitalizations (HFH) or | mITT Population |
| | 14.2.1.1.3 | all-cause mortalities, stratified by heart failure | i iiii i i opulation |
| | | ejection fraction | |
| <u> </u> | | ojootion naotion | L |

| | Table | | |
|---|---|---|---|
| Header | Number | Name | Analysis Set |
| | 14.2.1.1.3a | SAS-Output: 6-month incidence of HF | mITT Population |
| | | hospitalizations (HFH) or all-cause mortalities, | |
| | | stratified by heart failure ejection fraction | |
| | 14.2.1.1.4 | 6-month incidence of HF hospitalizations (HFH) or | Per Protocol |
| | | all-cause mortalities | Population |
| | 14.2.1.1.4a | SAS-Output: 6-month incidence of HF | Per Protocol |
| | 110115 | hospitalizations (HFH) or all-cause mortalities | Population |
| | 14.2.1.1.5 | 6-month incidence of HF hospitalizations (HFH) or | Cohort #1 |
| | 440445 | all-cause mortalities | Population |
| | 14.2.1.1.5a | SAS-Output: 6-month incidence of HF | Cohort #1 |
| | 110110 | hospitalizations (HFH) or all-cause mortalities | Population |
| | 14.2.1.1.6 | 6-month incidence of HF hospitalizations (HFH) or | mITT Population |
| | 14.2.1.1.6a | all-cause mortalities from CEC adjudication results | mITT Denulation |
| | 14.2.1.1.0a | SAS-Output: 6-month incidence of HF hospitalizations (HFH) or all-cause mortalities from | mITT Population |
| | | CEC adjudication results | |
| | 14.2.1.1.7 | 6-month incidence of HF hospitalizations (HFH) or | mITT Population |
| | | all-cause mortalities from CEC adjudication results, | opalation |
| | | stratified by sex | |
| | 14.2.1.1.7a | SAS-Output: 6-month incidence of HF | mITT Population |
| | | hospitalizations (HFH) or all-cause mortalities from | · |
| | | CEC adjudication results, stratified by sex | |
| | 14.2.1.1.8 | 6-month incidence of HF hospitalizations (HFH) or | mITT Population |
| | | all-cause mortalities from CEC adjudication results, | , |
| | | stratified by heart failure ejection fraction | |
| | 14.2.1.1.8a | SAS-Output: 6-month incidence of HF | mITT Population |
| | | hospitalizations (HFH) or all-cause mortalities from | |
| | | CEC adjudication results, stratified by heart failure | |
| | | ejection fraction | |
| | 14.2.1.1.9 | 6-month incidence of HF hospitalizations (HFH) or | Per Protocol |
| | 440440 | all-cause mortalities from CEC adjudication results | Population |
| | 14.2.1.1.9a | SAS-Output: 6-month incidence of HF | Per Protocol |
| | | hospitalizations (HFH) or all-cause mortalities from | Population |
| | 14.2.1.1.10 | CEC adjudication results | Cohort #1 |
| | 14.2.1.1.10 | 6-month incidence of HF hospitalizations (HFH) or all-cause mortalities from CEC adjudication results | |
| - | 14.2.1.1.10a | SAS-Output: 6-month incidence of HF | Population<br>Cohort #1 |
| | 17.2.1.1.100 | hospitalizations (HFH) or all-cause mortalities from | Population |
| | | CEC adjudication results | |
| | 14.2.1.1.11 | 6-month incidence of HF hospitalizations (HFH) | mITT Population |
| | | from CEC adjudication results | opalation |
| | 14.2.1.1.11a | SAS-Output: 6-month incidence of HF | mITT Population |
| | | hospitalizations (HFH) from CEC adjudication | ' |
| | | results | |
| | 14.2.1.1.12 | 6-month incidence of all-cause mortalities from CEC | mITT Population |
| | <u> </u> | adjudication results | <u>'</u> |
| | 14.2.1.1.12a | SÁS-Output: 6-month all-cause mortalities from | mITT Population |
| | | CEC adjudication results | • |
| | 14.2.1.2.2 | Sensitivity Analysis - 6-month incidence of HF | mITT Population |
| | | hospitalizations (HFH) or all-cause mortalities from | |
| | | CEC adjudication results using negative binomial | |
| | | regression model | |

SAP Version: 3.0 dated 17-Aug-2023 Controlled Document ID: **3903A.01**, Effective Date 29-Oct-2018 Filing requirements: TMF

| | Table | | |
|---|---|---|---|
| Header | Number | Name | Analysis Set |
| 110000 | 14.2.1.2.2a | SAS-Output: Sensitivity Analysis - 6-month | mITT Population |
| | | incidence of HF hospitalizations (HFH) or all-cause | ' |
| | | mortalities from CEC adjudication results using | |
| | | negative binomial regression model | |
| 14.2.2 | | Secondary Efficacy Parameters | |
| 14.2.2.1 | | Incidence of HF Hospitalizations or all-cause | |
| | | mortality at 12 months | |
| | 14.2.2.1.1 | 12-month incidence of HF hospitalizations (HFH) or | mITT Population |
| | | all-cause mortalities | · |
| | 14.2.2.1.1a | SAS-Output: 12-month incidence of HF | mITT Population |
| | | hospitalizations (HFH) or all-cause mortalities | |
| | 14.2.2.1.2 | 12-month incidence of HF hospitalizations (HFH) or | mITT Population |
| | | all-cause mortalities, stratified by sex | |
| | 14.2.2.1.2a | SAS-Output: 12-month incidence of HF | mITT Population |
| | | hospitalizations (HFH) or all-cause mortalities, | |
| | | stratified by sex | <u> </u> |
| | 14.2.2.1.3 | 12-month incidence of HF hospitalizations (HFH) or | mITT Population |
| | | all-cause mortalities, stratified by heart failure | |
| | | ejection fraction | |
| | 14.2.2.1.3a | SAS-Output: 12-month incidence of HF | mITT Population |
| | | hospitalizations (HFH) or all-cause mortalities, | |
| | 110011 | stratified by heart failure ejection fraction | <u> </u> |
| | 14.2.2.1.4 | 12-month incidence of HF hospitalizations (HFH) or | Per Protocol |
| | 110011 | all-cause mortalities | Population |
| | 14.2.2.1.4a | SAS-Output: 12-month incidence of HF | Per Protocol |
| | 14 2 2 4 5 | hospitalizations (HFH) or all-cause mortalities | Population<br>Cohort #1 |
| | 14.2.2.1.5 | 12-month incidence of HF hospitalizations (HFH) or all-cause mortalities | |
| | 14.2.2.1.5a | SAS-Output:12-month incidence of HF | Population<br>Cohort #1 |
| | 14.2.2.1.Ja | hospitalizations (HFH) or all-cause mortalities | Population |
| | 14.2.2.1.6 | Sensitivity Analysis - 12-month incidence of HF | mITT Population |
| | 14.2.2.1.0 | hospitalizations (HFH) or all-cause mortalities using | |
| | | negative binomial regression model | |
| | 14.2.2.1.6a | SAS-Output: Sensitivity Analysis - 12-month | mITT Population |
| | | incidence of HF hospitalizations (HFH) or all-cause | |
| | | mortalities using negative binomial regression | |
| | | model | |
| | 14.2.2.1.7 | 12-month incidence of HF hospitalizations (HFH) or | mITT Population |
| | | all-cause mortalities from CEC adjudication results | ·<br> |
| | 14.2.2.1.7a | SAS-Output: 12-month incidence of HF | mITT Population |
| | | hospitalizations (HFH) or all-cause mortalities from | |
| | | CEC adjudication results | |
| | 14.2.2.1.8 | 12-month incidence of HF hospitalizations (HFH) or | mITT Population |
| | | all-cause mortalities from CEC adjudication results, | |
| | | stratified by sex | |
| | 14.2.2.1.8a | SAS-Output: 12-month incidence of HF | mITT Population |
| | | hospitalizations (HFH) or all-cause mortalities from | |
| | | CEC adjudication results, stratified by sex | |
| | 14.2.2.1.9 | 12-month incidence of HF hospitalizations (HFH) or | mITT Population |
| | | all-cause mortalities from CEC adjudication results, | |
| | <u> </u> | stratified by heart failure ejection fraction | |

| | Table | | |
|---|---|---|---|
| Header | Number | Name | Analysis Set |
| | 14.2.2.1.9a | SAS-Output: 12-month incidence of HF | mITT Population |
| | | hospitalizations (HFH) or all-cause mortalities from | |
| | | CEC adjudication results, stratified by heart failure | |
| | 14.2.2.1.10 | ejection fraction 12-month incidence of HF hospitalizations (HFH) or | Per Protocol |
| | 14.2.2.1.10 | all-cause mortalities from CEC adjudication results | Population |
| | 14.2.2.1.10a | SAS-Output: 12-month incidence of HF | Per Protocol |
| | | hospitalizations (HFH) or all-cause mortalities from | Population |
| | | CEĊ adjudication results | ' |
| | 14.2.2.1.11 | 12-month incidence of HF hospitalizations (HFH) or | Cohort #1 |
| | | all-cause mortalities from CEC adjudication results | Population |
| | 14.2.2.1.11a | SAS-Output:12-month incidence of HF | Cohort #1 |
| | | hospitalizations (HFH) or all-cause mortalities from CEC adjudication results | Population |
| | 14.2.2.1.12 | Sensitivity Analysis - 12-month incidence of HF | mITT Population |
| | | hospitalizations (HFH) or all-cause mortalities from | |
| | | CEC adjudication results using negative binomial | |
| | 14.2.2.1.12a | regression model SAS-Output: Sensitivity Analysis - 12-month | mITT Population |
| | 14.2.2.1.12α | incidence of HF hospitalizations (HFH) or all-cause | |
| | | mortalities from CEC adjudication results using | |
| | | negative binomial regression model | |
| 14.2.2.2 | | Number of HF Hospitalizations at 6 and 12 months | |
| | | post-implant compared to the number of HF | |
| | | Hospitalizations in the 6 and 12 months prior to | |
| | 110001 | implant | |
| | 14.2.2.2.1 | Number of pre and post implant HF hospitalizations at 6 and 12 months post implant visit | mITT Population |
| | 14.2.2.2.2 | Number of pre and post implant HF hospitalizations | mITT Population |
| | 17.2.2.2.2 | at 6 and 12 months post implant visit, stratified by | |
| | | sex | |
| | 14.2.2.2.3 | Number of pre and post implant HF hospitalizations | mITT Population |
| | | at 6 and 12 months post implant visit, stratified by | |
| | | heart failure ejection fraction | |
| | 14.2.2.2.4 | Number of pre and post implant HF hospitalizations | Per Protocol |
| | 140005 | at 6 and 12 months post implant visit | Population |
| | 14.2.2.2.5 | Number of pre and post implant HF hospitalizations at 6 and 12 months post implant visit | Cohort #1<br>Population |
| | 14.2.2.2.6 | Number of pre and post implant HF hospitalizations | mITT Population |
| | 17.2.2.2.0 | at 6 and 12 months post implant visit from CEC | Thirt i opulation |
| | | adjudication results | |
| | 14.2.2.2.7 | Number of pre and post implant HF hospitalizations | mITT Population |
| | | at 6 and 12 months post implant visit from CEC | |
| | | adjudication results, stratified by sex | |
| | 14.2.2.2.8 | Number of pre and post implant HF hospitalizations | mITT Population |
| | | at 6 and 12 months post implant visit from CEC | |
| | | adjudication results, stratified by heart failure | |
| | 14.2.2.2.9 | ejection fraction Number of pre and post implant HF hospitalizations | Per Protocol |
| | 14.2.2.2.3 | at 6 and 12 months post implant visit from CEC | Population |
| | | adjudication results | . 500,000 |
| | 1 | aajaaloaton loodito | 1 |

| | Table | | |
|---|---|---|---|
| Header | Number | Name | Analysis Set |
| | 14.2.2.2.10 | Number of pre and post implant HF hospitalizations | Cohort #1 |
| | | at 6 and 12 months post implant visit from CEC | Population |
| | | adjudication results | |
| 14.2.2.3 | | Comparison of the number of HF Hospitalizations or | |
| | | Emergency Department/ Hospital Outpatient IV | |
| | | diuretic visits of Cohort #1 and Cohort #2 + Cohort | |
| | 110001 | #3 at 6 and 12 months post implant | |
| | 14.2.2.3.1 | Comparison of HF hospitalizations or HF | Comparison |
| | | emergency department/hospital outpatient IV | population |
| | | diuretic visits of Cohort #1 and Cohort #2 + Cohort | |
| | 14.2.2.3.1a | #3 at 6 and 12 months post implant visit | Comparison |
| | 14.2.2.3.1a | SAS-Output: Comparison of HF hospitalizations or HF emergency department/hospital outpatient IV | Comparison population |
| | | diuretic visits of Cohort #1 and Cohort #2 + Cohort | population |
| | | #3 at 6 and 12 months post implant visit | |
| | 14.2.2.3.2 | Comparison of HF hospitalizations or HF | Comparison |
| | 17.2.2.0.2 | emergency department/hospital outpatient IV | population |
| | | diuretic visits of Cohort #1 and Cohort #2 + Cohort | Population |
| | | #3 at 6 and 12 months post implant visit, stratified | |
| | | by sex | |
| | 14.2.2.3.2a | SAS-Output: Comparison of HF hospitalizations or | Comparison |
| | | HF emergency department/hospital outpatient IV | population |
| | | diuretic visits of Cohort #1 and Cohort #2 + Cohort | ' ' |
| | | #3 at 6 and 12 months post implant visit, stratified | |
| | | by sex | |
| | 14.2.2.3.3 | Comparison of HF hospitalizations or HF | Comparison |
| | | emergency department/hospital outpatient IV | population |
| | | diuretic visits of Cohort #1 and Cohort #2 + Cohort | |
| | | #3 at 6 and 12 months post implant visit, stratified | |
| | | by heart failure ejection fraction | _ |
| | 14.2.2.3.3a | SAS-Output: Comparison of HF hospitalizations or | Comparison |
| | | HF emergency department/hospital outpatient IV | population |
| | | diuretic visits of Cohort #1 and Cohort #2 + Cohort | |
| | | #3 at 6 and 12 months post implant visit, stratified | |
| | 140004 | by heart failure ejection fraction | Companies |
| | 14.2.2.3.4 | Comparison of HF hospitalizations or HF emergency department/hospital outpatient IV | Comparison |
| | | diuretic visits of Cohort #1 and Cohort #2 + Cohort | population |
| | | #3 at 6 and 12 months post implant visit from CEC | |
| | | adjudication results | |
| | 14.2.2.3.4a | SAS-Output: Comparison of HF hospitalizations or | Comparison |
| | 17.2.2.3.40 | HF emergency department/hospital outpatient IV | population |
| | | diuretic visits of Cohort #1 and Cohort #2 + Cohort | Population |
| | | #3 at 6 and 12 months post implant visit from CEC | |
| | | adjudication results | |
| | 14.2.2.3.5 | Comparison of HF hospitalizations or HF | Comparison |
| | | emergency department/hospital outpatient IV | population |
| | | diuretic visits of Cohort #1 and Cohort #2 + Cohort | ' |
| | | #3 at 6 and 12 months post implant visit from CEC | |
| | | adjudication results, stratified by sex | |

| | Table | | |
|---|---|---|---|
| Header | Number | Name | Analysis Set |
| | 14.2.2.3.5a | SAS-Output: Comparison of HF hospitalizations or HF emergency department/hospital outpatient IV diuretic visits of Cohort #1 and Cohort #2 + Cohort #3 at 6 and 12 months post implant visit from CEC adjudication results, stratified by sex | Comparison<br>population |
| | 14.2.2.3.6 | Comparison of HF hospitalizations or HF emergency department/hospital outpatient IV diuretic visits of Cohort #1 and Cohort #2 + Cohort #3 at 6 and 12 months post implant visit from CEC adjudication results, stratified by heart failure ejection fraction | Comparison<br>population |
| | 14.2.2.3.6a | SAS-Output: Comparison of HF hospitalizations or HF emergency department/hospital outpatient IV diuretic visits of Cohort #1 and Cohort #2 + Cohort #3 at 6 and 12 months post implant visit from CEC adjudication results, stratified by heart failure ejection fraction | Comparison<br>population |
| 14.2.2.4 | | Change of N-terminal pro B-type Natriuretic Peptide (NT-pro BNP) from Baseline through 6 and 12 months | |
| | 14.2.2.4.1 | NT-proBNP: summary by visit and change from baseline through 12 months | mITT Population |
| | 14.2.2.4.2 | NT-proBNP: summary by visit and change from baseline through 12 months, stratified by sex | mITT Population |
| | 14.2.2.4.3 | NT-proBNP: summary by visit and change from baseline through 12 months, stratified by heart failure ejection fraction | mITT Population |
| | 14.2.2.4.4 | NT-proBNP: summary by visit and change from baseline through 12 months | Per Protocol Population |
| | 14.2.2.4.5 | NT-proBNP: summary by visit and change from baseline through 12 months | Cohort #1<br>Population |
| 14.2.2.5 | | Combined outcome of a. First and recurrent HF Hospitalizations b. Emergency Department/ Hospital Outpatient IV diuretic visits c. all-cause mortality at 6 months, added together with equal weighting into a total number of events. | |
| | 14.2.2.5.1 | Number of events resulted from HF hospitalizations, HF emergency department/hospital outpatient IV diuretic visits and all-cause mortality at 6 months post implant visit | mITT Population |
| | 14.2.2.5.2 | Number of events resulted from HF hospitalizations, HF emergency department/hospital outpatient IV diuretic visits and all-cause mortality at 6 months post implant visit, stratified by sex | mITT Population |
| | 14.2.2.5.3 | Number of events resulted from HF hospitalizations, HF emergency department/hospital outpatient IV diuretic visits and all-cause mortality at 6 months post implant visit, stratified by heart failure ejection fraction | mITT Population |

| | Table | | |
|---|---|---|---|
| Header | Number | Name | Analysis Set |
| | 14.2.2.5.4 | Number of events resulted from HF hospitalizations, HF emergency department/hospital outpatient IV diuretic visits and all-cause mortality at 6 months post implant visit | Per Protocol<br>Population |
| | 14.2.2.5.5 | Number of events resulted from HF hospitalizations, HF emergency department/hospital outpatient IV diuretic visits and all-cause mortality at 6 months post implant visit | Cohort #1<br>Population |
| | 14.2.2.5.6 | Number of events resulted from HF hospitalizations, HF emergency department/hospital outpatient IV diuretic visits and all-cause mortality at 6 months post implant visit from CEC adjudication results | mITT Population |
| | 14.2.2.5.7 | Number of events resulted from HF hospitalizations, HF emergency department/hospital outpatient IV diuretic visits and all-cause mortality at 6 months post implant visit from CEC adjudication results, stratified by sex | mlTT Population |
| | 14.2.2.5.8 | Number of events resulted from HF hospitalizations, HF emergency department/hospital outpatient IV diuretic visits and all-cause mortality at 6 months post implant visit from CEC adjudication results, stratified by heart failure ejection fraction | mITT Population |
| | 14.2.2.5.9 | Number of events resulted from HF hospitalizations, HF emergency department/hospital outpatient IV diuretic visits and all-cause mortality at 6 months post implant visit from CEC adjudication results | Per Protocol<br>Population |
| | 14.2.2.5.10 | Number of events resulted from HF hospitalizations, HF emergency department/hospital outpatient IV diuretic visits and all-cause mortality at 6 months post implant visit from CEC adjudication results | Cohort #1<br>Population |
| 14.2.2.6 | | Heart failure hospitalization or Emergency Department / Hospital Outpatient IV diuretic visits at 6 and 12 months | |
| | 14.2.2.6.1 | Number of events resulted from HF hospitalizations or HF emergency department/hospital outpatient IV diuretic visits at 6 and 12 months post implant visit | mITT Population |
| | 14.2.2.6.2 | Number of events resulted from HF hospitalizations or HF emergency department/hospital outpatient IV diuretic visits at 6 and 12 months post implant visit, stratified by sex | mITT Population |
| | 14.2.2.6.3 | Number of events resulted from HF hospitalizations or HF emergency department/hospital outpatient IV diuretic visits at 6 and 12 months post implant visit, stratified by heart failure ejection fraction | mITT Population |
| | 14.2.2.6.4 | Number of events resulted from HF hospitalizations or HF emergency department/hospital outpatient IV diuretic visits at 6 and 12 months post implant visit | Per Protocol<br>Population |
| | 14.2.2.6.5 | Number of events resulted from HF hospitalizations or HF emergency department/hospital outpatient IV diuretic visits at 6 and 12 months post implant visit | Cohort #1<br>Population |
| | 14.2.2.6.6 | Time to first heart failure hospitalization: Kaplan-<br>Meier | mITT Population |

| | Table | | |
|---|---|---|---|
| Header | Number | Name | Analysis Set |
| | 14.2.2.6.7 | Time to first heart failure hospitalization: Kaplan-<br>Meier, stratified by sex | mITT Population |
| | 14.2.2.6.8 | Time to first heart failure hospitalization: Kaplan-<br>Meier, stratified by heart failure ejection fraction | mITT Population |
| | 14.2.2.6.9 | Time to first heart failure hospitalization: Kaplan-<br>Meier | Per Protocol<br>Population |
| | 14.2.2.6.10 | Time to first heart failure hospitalization: Kaplan-<br>Meier | Cohort #1<br>Population |
| | 14.2.2.6.11 | Time to first heart failure emergency department/hospital outpatient IV diuretic visit: Kaplan-Meier | mITT Population |
| | 14.2.2.6.12 | Time to first heart failure emergency department/hospital outpatient IV diuretic visit: Kaplan-Meier, stratified by sex | mITT Population |
| | 14.2.2.6.13 | Time to first heart failure emergency department/hospital outpatient IV diuretic visit: Kaplan-Meier, stratified by heart failure ejection fraction | mITT Population |
| | 14.2.2.6.14 | Time to first heart failure emergency department/hospital outpatient IV diuretic visit: Kaplan-Meier | Per Protocol<br>Population |
| | 14.2.2.6.15 | Time to first heart failure emergency department/hospital outpatient IV diuretic visit: Kaplan-Meier | Cohort #1<br>Population |
| | 14.2.2.6.26 | Number of events resulted from HF hospitalizations or HF emergency department/hospital outpatient IV diuretic visits at 6 and 12 months post implant visit from CEC adjudication results | mITT Population |
| | 14.2.2.6.27 | Number of events resulted from HF hospitalizations or HF emergency department/hospital outpatient IV diuretic visits at 6 and 12 months post implant visit from CEC adjudication results, stratified by sex | mITT Population |
| | 14.2.2.6.28 | Number of events resulted from HF hospitalizations or HF emergency department/hospital outpatient IV diuretic visits at 6 and 12 months post implant visit from CEC adjudication results, stratified by heart failure ejection fraction | mITT Population |
| | 14.2.2.6.29 | Number of events resulted from HF hospitalizations or HF emergency department/hospital outpatient IV diuretic visits at 6 and 12 months post implant visit from CEC adjudication results | Per Protocol<br>Population |
| | 14.2.2.6.30 | Number of events resulted from HF hospitalizations or HF emergency department/hospital outpatient IV diuretic visits at 6 and 12 months post implant visit from CEC adjudication results | Cohort #1<br>Population |
| | 14.2.2.6.31 | Time to first heart failure hospitalization from CEC adjudication results: Kaplan-Meier | mITT Population |
| | 14.2.2.6.32 | Time to first heart failure hospitalization from CEC adjudication results: Kaplan-Meier, stratified by sex | mITT Population |
| | 14.2.2.6.33 | Time to first heart failure hospitalization from CEC adjudication results: Kaplan-Meier, stratified by heart failure ejection fraction | mITT Population |

SAP Version: 3.0 dated 17-Aug-2023 Controlled Document ID: **3903A.01**, Effective Date 29-Oct-2018 Filing requirements: TMF

| Table | | |
|---|---|---|
| Header Number Name | | Analysis Set |
| | ilure hospitalization from CEC | Per Protocol |
| adjudication results | | Population |
| | ilure hospitalization from CEC | Cohort #1 |
| adjudication results | | Population |
| 14.2.2.6.36 Time to first heart f | ailure emergency | mITT Population |
| | outpatient IV diuretic visit from | |
| | esults: Kaplan-Meier | 177 D. 1 (' |
| 14.2.2.6.37 Time to first heart f | | mITT Population |
| | outpatient IV diuretic visit from | |
| 1 1 - | sults: Kaplan-Meier, stratified by | |
| 14.2.2.6.38 Time to first heart f | ailura amarganay | mITT Population |
| | outpatient IV diuretic visit from | IIII I Fopulation |
| | sults: Kaplan-Meier, stratified by | |
| heart failure ejection | | |
| 14.2.2.6.39 Time to first heart f | | Per Protocol |
| | outpatient IV diuretic visit from | Population |
| | esults: Kaplan-Meier | • |
| 14.2.2.6.40 Time to first heart f | ailure emergency | Cohort #1 |
| | outpatient IV diuretic visit from | Population |
| | esults: Kaplan-Meier | |
| 14.2.2.7 Cardiac and all-cau | | |
| I I | l all-cause mortality: Kaplan- | mITT Population |
| Meier | | ITT D ' '' |
| | l all-cause mortality: Kaplan- | mITT Population |
| Meier, stratified by 14.2.2.7.3 Time to cardiac and | sex<br>I all-cause mortality: Kaplan- | mITT Population |
| | heart failure ejection fraction | mini Fupulation |
| | I all-cause mortality: Kaplan- | Per Protocol |
| Meier | saass mortanty. Rapidit | Population |
| | l all-cause mortality: Kaplan- | Cohort #1 |
| Meier | | Population |
| | all-cause mortality from CEC | mITT Population |
| adjudication results | : Kaplan-Meier | • |
| | all-cause mortality from CEC | mITT Population |
| | Kaplan-Meier, stratified by sex | |
| | all-cause mortality from CEC | mITT Population |
| | : Kaplan-Meier, stratified by | |
| heart failure ejection | | D D |
| | all-cause mortality from CEC | Per Protocol |
| adjudication results | | Population Cohort #1 |
| 14.2.2.7.20 Time to cardiac and adjudication results | all-cause mortality from CEC | Population |
| | of Hospital (DAOH) | ι οραιατιστί |
| | of Hospital (DAOH) at 6 and 12 | mITT Population |
| months post implai | | min i opulation |
| | of hospital (DAOH) at 6 and 12 | mITT Population |
| | nt visit, stratified by sex | opalation |
| | of hospital (DAOH) at 6 and 12 | mITT Population |
| | visit, stratified by heart failure | ' |
| ejection fraction | | |

| | Table | | |
|---|---|---|---|
| | Number | Name | Analysis Set |
| | 14.2.2.8.4 | Days alive and out of hospital (DAOH) at 6 and 12 | Per Protocol |
| | 440005 | months post implant visit | Population |
| | 14.2.2.8.5 | Days alive and out of hospital (DAOH) at 6 and 12 | Cohort #1 |
| 14 2 2 0 | | months post implant visit | Population |
| 14.2.2.9 | 14.2.2.9.1 | Intravenous (IV) diuretic visits Number of events resulted from hospital outpatient | mITT Donulation |
| | 14.2.2.9.1 | IV diuretic visits at 6 and 12 months post implant | mITT Population |
| | | Visit | |
| | 14.2.2.9.2 | Number of events resulted from hospital outpatient | mITT Population |
| | | IV diuretic visits at 6 and 12 months post implant | |
| | | visit, stratified by sex | |
| | 14.2.2.9.3 | Number of events resulted from hospital outpatient | mITT Population |
| | | IV diuretic visits at 6 and 12 months post implant | |
| | | visit, stratified by heart failure ejection fraction | |
| | 14.2.2.9.4 | Number of events resulted from hospital outpatient | Per Protocol |
| | | IV diuretic visits at 6 and 12 months post implant | Population |
| <b>—</b> | 44000 | visit | 0-1 |
| | 14.2.2.9.5 | Number of events resulted from hospital outpatient | Cohort #1 |
| | | IV diuretic visits at 6 and 12 months post implant visit | Population |
| | 14.2.2.9.6 | Number of events resulted from hospital outpatient | mITT Population |
| | 14.2.2.9.0 | IV diuretic visits at 6 and 12 months post implant | illii i opulation |
| | | visit from CEC adjudication results | |
| | 14.2.2.9.7 | Number of events resulted from hospital outpatient | mITT Population |
| | | IV diuretic visits at 6 and 12 months post implant | ' |
| | | visit from CEC adjudication results, stratified by sex | |
| | 14.2.2.9.8 | Number of events resulted from hospital outpatient | mITT Population |
| | | IV diuretic visits at 6 and 12 months post implant | |
| | | visit from CEC adjudication results, stratified by | |
| | 14.2.2.9.9 | heart failure ejection fraction | Per Protocol |
| | 14.2.2.9.9 | Number of events resulted from hospital outpatient IV diuretic visits at 6 and 12 months post implant | Population |
| | | visit from CEC adjudication results | Fopulation |
| | 14.2.2.9.10 | Number of events resulted from hospital outpatient | Cohort #1 |
| | 14.2.2.0.10 | IV diuretic visits at 6 and 12 months post implant | Population |
| | | visit from CEC adjudication results | |
| 14.2.2.10 | | Heart failure related medication changes | |
| | 14.2.2.10.1 | Heart failure related medication changes by visits | mITT Population |
| | 14.2.2.10.2 | Heart failure related medication changes by visits, | mITT Population |
| | | stratified by sex | |
| | 14.2.2.10.3 | Heart failure related medication changes by visits, | mITT Population |
| <u> </u> | 44.0.0.40.4 | stratified by heart failure ejection fraction | Dan Danta I |
| | 14.2.2.10.4 | Heart failure related medication changes by visits | Per Protocol |
| <b>—</b> | 14 2 2 42 5 | Loop failure related medication shares a house it. | Population |
| | 14.2.2.10.5 | Heart failure related medication changes by visits | Cohort #1<br>Population |
| 14.2.2.11 | | Change in PA pressure | ι οραιατιστί |
| | 14.2.2.11.1 | Shifts in pulmonary artery pressure mean (mPAP) | mITT Population |
| | | classification from baseline to post-baseline visits | Spaidtion |
| | 14.2.2.11.2 | Shifts in pulmonary artery pressure mean (mPAP) | mITT Population |
| | | classification from baseline to post-baseline visits, | ' |
| | | stratified by sex | |

| | Table | | |
|---|---|---|---|
| Header | Number | Name | Analysis Set |
| | 14.2.2.11.3 | Shifts in pulmonary artery pressure mean (mPAP) classification from baseline to post-baseline visits, stratified by heart failure ejection fraction | mITT Population |
| | 14.2.2.11.4 | Shifts in pulmonary artery pressure mean (mPAP) classification from baseline to post-baseline visits | Per Protocol<br>Population |
| | 14.2.2.11.5 | Comparison between Cordella Sensor PA measurement before and after 6-Minute walk test by visit | mITT Population |
| | 14.2.2.11.6 | Comparison between Cordella Sensor PA measurement before and after 6-Minute walk test by visit, stratified by sex | mITT Population |
| | 14.2.2.11.7 | Comparison between Cordella Sensor PA measurement before and after 6-Minute walk test by visit, stratified by heart failure ejection fraction | mITT Population |
| | 14.2.2.11.8 | Comparison between Cordella Sensor PA measurement before and after 6-Minute walk test by visit | Per Protocol<br>Population |
| 14.2.2.12 | | Percentage of device success as documented by ability of the System to successfully transmit collected PAP data | |
| | 14.2.2.12.1 | Device success rate to transmit collected PAP data | mITT Population |
| | 14.2.2.12.2 | Device success rate to transmit collected PAP data | Per Protocol<br>Population |
| | 14.2.2.12.3 | Device success rate to transmit collected PAP data | Cohort #1<br>Population |
| 14.2.2.13 | | Quality of Life KCCQ questionnaire | |
| | 14.2.2.13.1 | Kansas City Cardiomyopathy Questionnaire (KCCQ): Summary for overall and domain scores by visit and change from baseline | mITT Population |
| | 14.2.2.13.2 | Kansas City Cardiomyopathy Questionnaire (KCCQ): Summary for overall and domain scores by visit and change from baseline | mITT Population |
| | 14.2.2.13.3 | Kansas City Cardiomyopathy Questionnaire (KCCQ): Summary for overall and domain scores by visit and change from baseline | mITT Population |
| | 14.2.2.13.4 | Kansas City Cardiomyopathy Questionnaire (KCCQ): Summary for overall and domain scores by visit and change from baseline | Per Protocol<br>Population |
| | 14.2.2.13.5 | Kansas City Cardiomyopathy Questionnaire (KCCQ): Summary for overall and domain scores by visit and change from baseline | Cohort #1<br>Population |
| 14.2.2.14 | | Functional status improvement | |
| | 14.2.2.14.1 | Shifts in NYHA functional classification from baseline to post-baseline visits | mITT Population |
| | 14.2.2.14.2 | Shifts in NYHA functional classification from baseline to post-baseline visits, stratified by sex | mITT Population |
| | 14.2.2.14.3 | Shifts in NYHA functional classification from baseline to post-baseline visits, stratified by heart failure ejection fraction | mITT Population |
| | 14.2.2.14.4 | Shifts in NYHA functional classification from baseline to post-baseline visits | Per Protocol<br>Population |

| | Table | | |
|---|---|---|---|
| Header | Number | Name | Analysis Set |
| | 14.2.2.14.5 | Shifts in NYHA functional classification from | Cohort #1 |
| | | baseline to post-baseline visits | Population |
| | 14.2.2.14.6 | Six (6)-Minute walk, summary by visit and change | mITT Population |
| | | from baseline | |
| | 14.2.2.14.7 | Six (6)-Minute walk, summary by visit and change from baseline, stratified by sex | mITT Population |
| | 14.2.2.14.8 | Six (6)-Minute walk, summary by visit and change from baseline, stratified by heart failure ejection fraction | mITT Population |
| | 14.2.2.14.9 | Six (6)-Minute walk, summary by visit and change from baseline | Per Protocol<br>Population |
| | 14.2.2.14.10 | Six (6)-Minute walk, summary by visit and change | Cohort #1 |
| | | from baseline | Population |
| 14.2.2.15 | | Supportive analysis to evaluate pooled site effect | |
| | 14.2.2.15.1 | Homogeneity test to evaluate of the pooled site effects | mITT Population |
| 14.3 | | Safety Data Summary Tables | |
| 14.3.1 | | Adverse Events | |
| 14.3.1.1 | | Primary Safety Endpoint | |
| | 14.3.1.1.1 | Freedom from device/system related complication at 6 months post implant visit | mITT Population |
| | 14.3.1.1.1a | SAS-Output: Freedom from device/system related complication at 6 months post implant visit | mITT Population |
| | 14.3.1.1.2 | Freedom from device/system related complication at 6 months post implant visit, stratified by sex | mITT Population |
| | 14.3.1.1.2a | SAS-Output: Freedom from device/system related complication at 6 months post implant visit, stratified by sex | mITT Population |
| | 14.3.1.1.3 | Freedom from device/system related complication at 6 months post implant visit, stratified by heart failure ejection fraction | mITT Population |
| | 14.3.1.1.3a | SAS-Output: Freedom from device/system related complication at 6 months post implant visit, stratified by heart failure ejection fraction | mITT Population |
| | 14.3.1.1.4.1 | Freedom from device/system related complication at 6 months post implant visit | Per Protocol Population |
| | 14.3.1.1.4.1 | SAS-Output: Freedom from device/system related | Per Protocol |
| | 14.3.1.1.4.2 | complication at 6 months post implant visit Freedom from device/system related complication at 6 months post implant visit | Population<br>ITT Population |
| | 14.3.1.1.4.2 | SAS-Output: Freedom from device/system related | ITT Population |
| | a<br>14.3.1.1.5a | complication at 6 months post implant visit SAS-Output: Freedom from device/system related | Cohort #1 |
| | | complication at 6 months post implant visit | Population |
| | 14.3.1.1.6 | Freedom from device/system related complication at 6 months post implant visit - Extreme cases sensitivity analysis | mITT Population |
| | 14.3.1.1.6a | SAS-Output: Freedom from device/system related complication at 6 months post implant visit - Extreme cases sensitivity analysis | mITT Population |

| | Table | | |
|---|---|---|---|
| Header | Number | Name | Analysis Set |
| | 14.3.1.1.7 | Freedom from device/system related complication at 12 months post implant visit - Tipping point sensitivity analysis | mITT Population |
| | 14.3.1.1.7a | SAS-Output: Freedom from device/system related complication at 12 months post implant visit - Tipping point sensitivity analysis | mITT Population |
| | 14.3.1.1.13 | Freedom from device/system related complication at 6 months post implant visit from CEC adjudication results | mITT Population |
| | 14.3.1.1.13a | SAS-Output: Freedom from device/system related complication at 6 months post implant visit from CEC adjudication results | mITT Population |
| | 14.3.1.1.14 | Freedom from device/system related complication at 6 months post implant visit from CEC adjudication results, stratified by sex | mITT Population |
| | 14.3.1.1.14a | SAS-Output: Freedom from device/system related complication at 6 months post implant visit from CEC adjudication results, stratified by sex | mITT Population |
| | 14.3.1.1.15 | Freedom from device/system related complication at 6 months post implant visit from CEC adjudication results, stratified by heart failure ejection fraction | mITT Population |
| | 14.3.1.1.15a | SAS-Output: Freedom from device/system related complication at 6 months post implant visit from CEC adjudication results, stratified by heart failure ejection fraction | mITT Population |
| | 14.3.1.1.16.<br>1 | Freedom from device/system related complication at 6 months post implant visit from CEC adjudication results | Per Protocol<br>Population |
| | 14.3.1.1.16.<br>1a | SAS-Output: Freedom from device/system related complication at 6 months post implant visit from CEC adjudication results | Per Protocol<br>Population |
| | 14.3.1.1.16.<br>2 | Freedom from device/system related complication at 6 months post implant visit from CEC adjudication results | ITT Population |
| | 14.3.1.1.16.<br>2a | SAS-Output: Freedom from device/system related complication at 6 months post implant visit from CEC adjudication results | ITT Population |
| | 14.3.1.1.17 | Freedom from device/system related complication at 6 months post implant visit from CEC adjudication results | Cohort #1<br>Population |
| | 14.3.1.1.17a | SAS-Output: Freedom from device/system related complication at 6 months post implant visit from CEC adjudication results | Cohort #1<br>Population |
| | 14.3.1.1.18 | Freedom from device/system related complication at 6 months post implant visit from CEC adjudication results - Extreme cases sensitivity analysis | mITT Population |
| | 14.3.1.1.18a | SAS-Output: Freedom from device/system related complication at 6 months post implant visit from CEC adjudication results - Extreme cases sensitivity analysis | mITT Population |

| | Table | | |
|---|---|---|---|
| Header | Number | Name | Analysis Set |
| | 14.3.1.1.19 | Freedom from device/system related complication at | mITT Population |
| | | 12 months post implant visit from CEC adjudication | |
| | | results - Tipping point sensitivity analysis | |
| | 14.3.1.1.19a | SAS-Output: Freedom from device/system related | mITT Population |
| | | complication at 12 months post implant visit from | |
| | | CEC adjudication results - Tipping point sensitivity | |
| | 14.3.1.2.1 | analysis | mITT Denulation |
| | 14.3.1.2.1 | Freedom from pressure sensor failure at 6 months post implant visit | mITT Population |
| | 14.3.1.2.1a | SAS-Output: Freedom from pressure sensor failure | mITT Population |
| | 14.0.1.2.14 | at 6 months post implant visit | |
| | 14.3.1.2.2 | Freedom from pressure sensor failure at 6 months | mITT Population |
| | 1 1101 11212 | post implant visit, stratified by sex | Time to paration |
| | 14.3.1.2.2a | SAS-Output: Freedom from pressure sensor failure | mITT Population |
| | | at 6 months post implant visit, stratified by sex | |
| | 14.3.1.2.3 | Freedom from pressure sensor failure at 6 months | mITT Population |
| | | post implant visit, stratified by heart failure ejection | |
| | | fraction | |
| | 14.3.1.2.3a | SAS-Output: Freedom from pressure sensor failure | mITT Population |
| | | at 6 months post implant visit, stratified by heart | |
| | 4404044 | failure ejection fraction | Day Dyata and |
| | 14.3.1.2.4.1 | Freedom from pressure sensor failure at 6 months | Per Protocol |
| | 14.3.1.2.4.1 | post implant visit SAS-Output: Freedom from pressure sensor failure | Population Per Protocol |
| | a | at 6 months post implant visit | Population |
| | 14.3.1.2.4.2 | Freedom from pressure sensor failure at 6 months | ITT Population |
| | 1 1.0. 1.2. 1.2 | post implant visit | TTTT Opalation |
| | 14.3.1.2.4.2 | SAS-Output: Freedom from pressure sensor failure | ITT Population |
| | а | at 6 months post implant visit | • |
| | 14.3.1.2.5a | SAS-Output: Freedom from pressure sensor failure | Cohort #1 |
| | | at 6 months post implant visit | Population |
| | 14.3.1.2.6 | Freedom from pressure sensor failure at 6 months | mITT Population |
| | | post implant visit - Extreme cases sensitivity | |
| | 14 2 4 2 2 - | analysis | mITT Demilation |
| | 14.3.1.2.6a | SAS-Output: Freedom from pressure sensor failure | mITT Population |
| | | at 6 months post implant visit - Extreme cases sensitivity analysis | |
| | 14.3.1.2.7 | Freedom from pressure sensor failure at 6 months | mITT Population |
| | 1 | post implant visit - Tipping point sensitivity analysis | Opalation |
| | 14.3.1.2.7a | SAS-Output: Freedom from pressure sensor failure | mITT Population |
| | | at 6 months post implant visit - Tipping point | |
| | | sensitivity analysis | |
| | 14.3.1.2.13 | Freedom from pressure sensor failure at 6 months | mITT Population |
| | | post implant visit from CEC adjudication results | |
| | 14.3.1.2.13a | SAS-Output: Freedom from pressure sensor failure | mITT Population |
| | | at 6 months post implant visit from CEC adjudication | |
| | 1110101 | results | |
| | 14.3.1.2.14 | Freedom from pressure sensor failure at 6 months | mITT Population |
| | | post implant visit from CEC adjudication results, | |
| | <u> </u> | stratified by sex | |

| | Table | | |
|---|---|---|---|
| Header | Number | Name | Analysis Set |
| | 14.3.1.2.14a | SAS-Output: Freedom from pressure sensor failure | mITT Population |
| | | at 6 months post implant visit from CEC adjudication | |
| | | results, stratified by sex | |
| | 14.3.1.2.15 | Freedom from pressure sensor failure at 6 months | mITT Population |
| | | post implant visit from CEC adjudication results, | |
| | 14.0.4.0.45- | stratified by heart failure ejection fraction | molTT Demodetien |
| | 14.3.1.2.15a | SAS-Output: Freedom from pressure sensor failure | mITT Population |
| | | at 6 months post implant visit from CEC adjudication results, stratified by heart failure ejection fraction | |
| | 14.3.1.2.16. | Freedom from pressure sensor failure at 6 months | Per Protocol |
| | 14.0.1.2.10. | post implant visit from CEC adjudication results | Population |
| | 14.3.1.2.16. | SAS-Output: Freedom from pressure sensor failure | Per Protocol |
| | 1a | at 6 months post implant visit from CEC adjudication | Population |
| | | results | |
| | 14.3.1.2.16. | Freedom from pressure sensor failure at 6 months | ITT Population |
| | 2 | post implant visit from CEC adjudication results | · |
| | 14.3.1.2.16. | SAS-Output: Freedom from pressure sensor failure | ITT Population |
| | 2a | at 6 months post implant visit from CEC adjudication | |
| | | results | |
| | 14.3.1.2.17a | SAS-Output: Freedom from pressure sensor failure | Cohort #1 |
| | | at 6 months post implant visit from CEC adjudication | Population |
| | 14 2 4 2 40 | results | mITT Denulation |
| | 14.3.1.2.18 | Freedom from pressure sensor failure at 6 months post implant visit from CEC adjudication results - | mITT Population |
| | | Extreme cases sensitivity analysis | |
| | 14.3.1.2.18a | SAS-Output: Freedom from pressure sensor failure | mITT Population |
| | 11.0.1.2.104 | at 6 months post implant visit from CEC adjudication | IIII Opalation |
| | | results - Extreme cases sensitivity analysis | |
| | 14.3.1.2.19 | Freedom from pressure sensor failure at 6 months | mITT Population |
| | | post implant visit from CEC adjudication results - | |
| | | Tipping point sensitivity analysis | |
| | 14.3.1.2.19a | SAS-Output: Freedom from pressure sensor failure | mITT Population |
| | | at 6 months post implant visit from CEC adjudication | |
| | 110101 | results - Tipping point sensitivity analysis | 177 D 1 (' |
| | 14.3.1.3.1 | Adverse events – Overall summary | ITT Population |
| | 14.3.1.3.2 | Adverse events – Overall summary, stratified by sex | |
| | 14.3.1.3.3 | Adverse events – Overall summary, stratified by | ITT Population |
| | 14.3.1.3.4 | heart failure ejection fraction | Por Protocol |
| | 14.3.1.3.4 | Adverse events – Overall summary | Per Protocol Population |
| | 14.3.1.3.5 | Adverse events – Overall summary | Cohort #1 |
| | 14.0.1.0.0 | Adverse events – Overall summary | Population |
| | 14.3.1.4.1 | Predefined adverse events by category | ITT Population |
| | 14.3.1.4.2 | Predefined adverse events by category, stratified | ITT Population |
| | | sex | |
| | 14.3.1.4.3 | Predefined adverse events by category, stratified by | ITT Population |
| | | heart failure ejection fraction | <u>'</u> |
| | 14.3.1.4.4 | Predefined adverse events by category | Per Protocol |
| | | | Population |
| | 14.3.1.4.5 | Predefined adverse events by category | Cohort #1 |
| | | | Population |

| | Table | | |
|---|---|---|---|
| Header | Number | Name | Analysis Set |
| | 14.3.1.5.1 | Adverse Events by System Organ Class and Preferred Term | ITT Population |
| | 14.3.1.5.2 | Adverse Events by System Organ Class and Preferred Term, stratified by sex | ITT Population |
| | 14.3.1.5.3 | Adverse Events by System Organ Class and Preferred Term, stratified by heart failure ejection fraction | ITT Population |
| | 14.3.1.5.4 | Adverse Events by System Organ Class and Preferred Term | Cohort #1<br>Population |
| | 14.3.1.6.1 | Serious Adverse Events by System Organ Class and Preferred Term | ITT Population |
| | 14.3.1.6.2 | Serious Adverse Events by System Organ Class and Preferred Term, stratified by sex | ITT Population |
| | 14.3.1.6.3 | Serious Adverse Events by System Organ Class and Preferred Term, stratified by heart failure ejection fraction | ITT Population |
| | 14.3.1.6.4 | Serious Adverse Events by System Organ Class and Preferred Term | Cohort #1<br>Population |
| | 14.3.1.7.1 | Serious Adverse Events by Preferred Term | ITT Population |
| | 14.3.1.7.2 | Serious Adverse Events by Preferred Term | Cohort #1<br>Population |
| | 14.3.1.8.1 | Serious Adverse Events by Seriousness Criteria | ITT Population |
| | 14.3.1.8.2 | Serious Adverse Events by Seriousness Criteria, stratified by sex | ITT Population |
| | 14.3.1.8.3 | Serious Adverse Events by Seriousness Criteria, stratified by heart failure ejection fraction | ITT Population |
| | 14.3.1.8.4 | Serious Adverse Events by Seriousness Criteria | Cohort #1<br>Population |
| | 14.3.1.9.1 | Serious Predefined Adverse Events by Category | ITT Population |
| | 14.3.1.9.2 | Serious Predefined Adverse Events by Category, stratified by sex | ITT Population |
| | 14.3.1.9.3 | Serious Predefined Adverse Events by Category, stratified by heart failure ejection fraction | ITT Population |
| | 14.3.1.9.4 | Serious Predefined Adverse Events by Category | Cohort #1<br>Population |
| | 14.3.1.10.1 | Study Procedure Related Adverse Events by System Organ Class and Preferred Term | ITT Population |
| | 14.3.1.10.2 | Study Procedure Related Adverse Events by<br>System Organ Class and Preferred Term | Cohort #1<br>Population |
| | 14.3.1.10.3 | Serious Study Procedure Related Adverse Events by System Organ Class and Preferred Term | ITT Population |
| | 14.3.1.10.4 | Serious Study Procedure Related Adverse Events by System Organ Class and Preferred Term | Cohort #1<br>Population |
| | 14.3.1.11.1 | Study Procedure Related Adverse Events by Procedure Type | ITT Population |
| | 14.3.1.11.2 | Study Procedure Related Adverse Events by Procedure Type | Cohort #1<br>Population |
| | 14.3.1.12.1 | Adverse Events by System Organ Class, Preferred Term, and Maximum Severity | ITT Population |
| | 14.3.1.12.2 | Adverse Events by System Organ Class, Preferred Term, and Maximum Severity | Cohort #1<br>Population |

| | Table | | |
|---|---|---|---|
| Header | Number | Name | Analysis Set |
| | 14.3.1.13.1 | Adverse Events by System Organ Class, Preferred | ITT Population |
| | | Term, and Maximum Relationship to Implant | - |
| | | Procedure | |
| | 14.3.1.13.2 | Adverse Events by System Organ Class, Preferred | Cohort #1 |
| | | Term, and Maximum Relationship to Implant | Population |
| | 110111 | Procedure | ITT Damidation |
| | 14.3.1.14.1 | Device/System-Related Complication by System | ITT Population |
| | 14.3.1.14.2 | Organ Class and Preferred Term Device/System-Related Complication by System | ITT Population |
| | 14.3.1.14.2 | Organ Class and Preferred Term, stratified by sex | III Population |
| | 14.3.1.14.3 | Device/System-Related Complication by System | ITT Population |
| | 1 1.0.1.11.0 | Organ Class and Preferred Term, stratified by heart | TTT T OPGIGNOTI |
| | | failure ejection fraction | |
| | 14.3.1.14.4 | Device/System-Related Complication by System | Cohort #1 |
| | | Organ Class and Preferred Term | Population |
| | 14.3.1.15.1 | Device/System-Related Complication by System | ITT Population |
| | | Organ Class, Preferred Term and Maximum | |
| | 1 1 2 1 1 5 5 | Severity | 0 1 1 "1 |
| | 14.3.1.15.2 | Device/System-Related Complication by System | Cohort #1 |
| | | Organ Class, Preferred Term and Maximum | Population |
| | 14 2 1 16 1 | Severity Device/System Related Complication by Revice | ITT Deputation |
| | 14.3.1.16.1<br>14.3.1.16.2 | Device/System-Related Complication by Device Device/System-Related Complication by Device | ITT Population Cohort #1 |
| | 14.3.1.10.2 | Device/System-Related Complication by Device | Population |
| | 14.3.1.17.1 | Unanticipated Adverse Device Effects by System | ITT Population |
| | 11.0.1.17.1 | Organ Class and Preferred Term | TTT T OPGIGNOTI |
| | 14.3.1.17.2 | Unanticipated Adverse Device Effects by System | Cohort #1 |
| | | Organ Class and Preferred Term | Population |
| | 14.3.1.18.1 | Unanticipated Adverse Device Effects by System | ITT Population |
| | | Organ Class, Preferred Term and Maximum | |
| | | Severity | |
| | 14.3.1.18.2 | Unanticipated Adverse Device Effects by System | Cohort #1 |
| | | Organ Class, Preferred Term and Maximum | Population |
| | 14 2 1 10 1 | Severity Unanticipated Adverse Device Effects by Device | ITT Deputation |
| | 14.3.1.19.1<br>14.3.1.19.2 | Unanticipated Adverse Device Effects by Device Unanticipated Adverse Device Effects by Device | |
| | 14.5.1.19.2 | Onanticipated Adverse Device Lifects by Device | Population |
| | 14.3.1.20.1 | Implant Procedure Related Adverse Events by | ITT Population |
| | 1 1.0. 1.20.1 | System Organ Class and Preferred Term | i opalation |
| | 14.3.1.20.2 | Implant Procedure Related Adverse Events by | Cohort #1 |
| | | System Organ Class and Preferred Term | Population |
| | 14.3.1.20.3 | Serious Implant Procedure Related Adverse Events | ITT Population |
| | | by System Organ Class and Preferred Term | |
| | 14.3.1.20.4 | Serious Implant Procedure Related Adverse Events | Cohort #1 |
| | 1440404 | by System Organ Class and Preferred Term | Population |
| | 14.3.1.21.1 | Predefined Adverse Events by Relationships to | ITT Population |
| | | Device and Study Procedure from CEC Adjudication | |
| | 14 2 1 21 2 | Results Prodefined Adverse Events by Poletionships to | Cobort #1 |
| | 14.3.1.21.2 | Predefined Adverse Events by Relationships to Device and Study Procedure from CEC Adjudication | Cohort #1<br>Population |
| | | Results | ι οραιαιιστί |
| | I . | Nosuito | |

| 1 | Number<br>14.3.1.22.1<br>14.3.1.22.2<br>14.3.1.23.1<br>14.3.1.23.2<br>14.3.1.24.1<br>14.3.1.24.2<br>14.3.1.25.1 | Name Adverse Events leading to Study Withdrawal by System Organ Class and Preferred Term Adverse Events leading to Study Withdrawal by System Organ Class and Preferred Term Device Deficiency Device Deficiency Pressure Sensor Failure AEs by System Organ Class and Preferred Term Pressure Sensor Failure AEs by System Organ Class and Preferred Term | Analysis Set ITT Population Cohort #1 Population ITT Population Cohort #1 Population ITT Population ITT Population |
|---|---|---|---|
| 1 | 14.3.1.22.2<br>14.3.1.23.1<br>14.3.1.23.2<br>14.3.1.24.1<br>14.3.1.24.2 | System Organ Class and Preferred Term Adverse Events leading to Study Withdrawal by System Organ Class and Preferred Term Device Deficiency Device Deficiency Pressure Sensor Failure AEs by System Organ Class and Preferred Term Pressure Sensor Failure AEs by System Organ | Cohort #1 Population ITT Population Cohort #1 Population |
| 1 | 14.3.1.23.1<br>14.3.1.23.2<br>14.3.1.24.1<br>14.3.1.24.2 | System Organ Class and Preferred Term Device Deficiency Device Deficiency Pressure Sensor Failure AEs by System Organ Class and Preferred Term Pressure Sensor Failure AEs by System Organ | Population ITT Population Cohort #1 Population |
| | 14.3.1.23.2<br>14.3.1.24.1<br>14.3.1.24.2 | Device Deficiency Device Deficiency Pressure Sensor Failure AEs by System Organ Class and Preferred Term Pressure Sensor Failure AEs by System Organ | ITT Population Cohort #1 Population |
| | 14.3.1.23.2<br>14.3.1.24.1<br>14.3.1.24.2 | Device Deficiency Pressure Sensor Failure AEs by System Organ Class and Preferred Term Pressure Sensor Failure AEs by System Organ | Cohort #1<br>Population |
| 1 | 14.3.1.24.1<br>14.3.1.24.2 | Pressure Sensor Failure AEs by System Organ Class and Preferred Term Pressure Sensor Failure AEs by System Organ | Population |
| | 14.3.1.24.2 | Class and Preferred Term Pressure Sensor Failure AEs by System Organ | |
| | 14.3.1.24.2 | Class and Preferred Term Pressure Sensor Failure AEs by System Organ | III Population |
| | | , , , | |
| | 14.3.1.25.1 | Class and Preferred Term | Cohort #1<br>Population |
| 1 | | Anticipated Adverse Events by System Organ Class and Preferred Term | ITT Population |
| 1 | 14.3.1.25.2 | Anticipated Adverse Events by System Organ Class | Cohort #1 |
| | | and Preferred Term | Population |
| | 14.3.1.26.1 | Anticipated Adverse Events by System Organ Class and Preferred Term and Maximum Severity | ITT Population |
| | 14.3.1.26.2 | Anticipated Adverse Events by System Organ Class and Preferred Term and Maximum Severity | Cohort #1<br>Population |
| 1 | 14.3.1.27.1 | Anticipated Adverse Events by System Organ Class and Preferred Term and Maximum Relationship to Implant Procedure | ITT Population |
| | 14.3.1.27.2 | Anticipated Adverse Events by System Organ Class and Preferred Term and Maximum Relationship to Implant Procedure | Cohort #1<br>Population |
| 1 | 14.3.1.28.1 | Unanticipated Adverse Events by System Organ Class and Preferred Term | ITT Population |
| 1 | 14.3.1.28.2 | Unanticipated Adverse Events by System Organ | Cohort #1 |
| <del> </del> | 14.3.1.29.1 | Class and Preferred Term | Population |
| | | Unanticipated Adverse Events by System Organ Class and Preferred Term and Maximum Severity | ITT Population |
| | 14.3.1.29.2 | Unanticipated Adverse Events by System Organ Class and Preferred Term and Maximum Severity | Cohort #1<br>Population |
| 1 | 14.3.1.30.1 | Unanticipated Adverse Events by System Organ Class and Preferred Term and Maximum Relationship to Implant Procedure | ITT Population |
| 1 | 14.3.1.30.2 | Unanticipated Adverse Events by System Organ<br>Class and Preferred Term and Maximum<br>Relationship to Implant Procedure | Cohort #1<br>Population |
| 1 | 14.3.1.31.1 | Other serious adverse events (AE) CEC adjudicated by system organ class and preferred term | ITT Population |
| | 14.3.1.31.2 | Other serious adverse events (AE) CEC adjudicated by system organ class and preferred term | Cohort #1<br>Population |
| 14.3.2 | | Listings of Deaths, Other Serious and Significant Adverse Events | |
| | 14.3.2.1.1 | Deaths from Adverse Event Page, Listing | Enrolled Population |
| | 14.3.2.1.2 | Deaths from Study Completion Page, Listing | Enrolled Population |
| | 14.3.2.1.3 | Deaths from Adverse Event Page, Listing | Cohort #1<br>Population |
| 1 | 14.3.2.1.4 | Deaths from Study Completion Page, Listing | Cohort #1<br>Population |
| 1 | 14.3.2.2 | Serious Adverse Events, Listing | Enrolled Population |

SAP Version: 3.0 dated 17-Aug-2023 Controlled Document ID: **3903A.01**, Effective Date 29-Oct-2018 Filing requirements: TMF

| | Table | | |
|---|---|---|---|
| Header | Number | Name | Analysis Set |
| | 14.3.2.3 | Unanticipated Adverse Device Effects, Listing | Enrolled Population |
| | 14.3.2.4 | Adverse Events Leading to Study Withdrawal, Listing | Enrolled Population |
| | 14.3.2.5 | Serious Adverse Events, Listing | Cohort #1<br>Population |
| | 14.3.2.6 | Unanticipated Adverse Device Effects, Listing | Cohort #1<br>Population |
| | 14.3.2.7 | Adverse Events Leading to Study Withdrawal, Listing | Cohort #1<br>Population |
| 14.3.3 | Not to be<br>used for any<br>Tables | Narratives of Deaths, Other Serious and Certain Other Significant Adverse Events | |
| 14.3.4 | | Abnormal Laboratory Value (each subject) | |
| 14.3.4.1 | | Clinical Laboratory Data | |
| 14.3.4.1.<br>1 | | Hematology Data | |
| | 14.3.4.1.1.1 | Hematology: Proportion of Abnormal Results by Visit | ITT Population |
| | 14.3.4.1.1.2 | Hematology: Abnormal Results, Listing | ITT Population |
| | 14.3.4.1.1.3 | Hematology: Proportion of Abnormal Results by Visit | Cohort #1<br>Population |
| | 14.3.4.1.1.4 | Hematology: Abnormal Results, Listing | Cohort #1 |
| | | | Population |
| 14.3.4.1.<br>2 | | Chemistry Data | |
| | 14.3.4.1.2.1 | Chemistry: Proportion of Abnormal Results by Visit | ITT Population |
| | 14.3.4.1.2.2 | Chemistry: Abnormal Results, Listing | ITT Population |
| | 14.3.4.1.2.3 | Chemistry: Proportion of Abnormal Results by Visit | Cohort #1<br>Population |
| | 14.3.4.1.2.4 | Chemistry: Abnormal Results, Listing | Cohort #1<br>Population |
| 14.3.4.1.<br>3 | | Urinalysis Data | |
| | 14.3.4.1.3.1 | Urinalysis: Proportion of Abnormal Results by Visit | |
| | 14.3.4.1.3.2 | Urinalysis: Abnormal Results, Listing | ITT Population |
| | 14.3.4.1.3.3 | Urinalysis: Proportion of Abnormal Results by Visit | Cohort #1 Population |
| | 14.3.4.1.3.4 | Urinalysis: Abnormal Results, Listing | Cohort #1<br>Population |
| 14.3.4.1.<br>4 | | Coagulation | |
| _ | 14.3.4.1.4.1 | Coagulation: Proportion of Abnormal Results by Visit | ITT Population |
| | 14.3.4.1.4.2 | Coagulation: Proportion of Abnormal Results by Visit | Cohort #1<br>Population |
| 14.3.4.1.<br>5 | | NT-pro BNP | |
| | 14.3.4.1.5.1 | NT-pro BNP: Proportion of Abnormal Results by Visit | ITT Population |
| | 14.3.4.1.5.2 | NT-pro BNP: Proportion of Abnormal Results by Visit | Cohort #1<br>Population |
| | Table | | |
|---|---|---|---|
| Header | Number | Name | Analysis Set |
| 14.3.4.2 | | Vital Signs | |
| | 14.3.4.2.1 | Vital Signs: Summary by Visit and Change from Baseline | ITT Population |
| | 14.3.4.2.1 | Vital Signs: Summary by Visit and Change from Baseline | Cohort #1<br>Population |
| 14.3.4.3 | | Electrocardiogram (ECG) Data | |
| | 14.3.4.3.1 | Summary of Overall ECG Evaluation by Visit | ITT Population |
| | 14.3.4.3.2 | Shift from Baseline of Overall ECG Evaluation to Each Visit | ITT Population |
| | 14.3.4.3.3 | Summary of Overall ECG Evaluation by Visit | Cohort #1<br>Population |
| | 14.3.4.3.4 | Shift from Baseline of Overall ECG Evaluation to Each Visit | Cohort #1<br>Population |
| 14.3.4.4 | | Echocardiogram Data | |
| | 14.3.4.4.1 | Summary of Overall Echocardiogram Evaluation by Visit | ITT Population |
| | 14.3.4.4.2 | Shift from Baseline of Overall Echocardiogram Evaluation to Each Visit | ITT Population |
| | 14.3.4.4.3 | Summary of Overall Echocardiogram Evaluation by Visit | Cohort #1<br>Population |
| | 14.3.4.4.4 | Shift from Baseline of Overall Echocardiogram Evaluation to Each Visit | Cohort #1<br>Population |
| 14.3.4.5 | | Physical Examination Results | |
| | 14.3.4.5.1 | Summary of Physical Examination Results at Screening | ITT Population |
| _ | 14.3.4.5.1 | Summary of Physical Examination Results at Screening | Cohort #1<br>Population |

# 15. Index of Figures

| Header | Table Number | Name | Analysis Set |
|---|---|---|---|
| 14.2 | | Efficacy Data Summary Figures and Tables | |
| 14.2.2 | | Secondary Efficacy Parameter | |
| | 14.2.2.6.16 | Time to first heart failure hospitalization: | mITT Population |
| | | Kaplan-Meier plot | |
| | 14.2.2.6.17 | Time to first heart failure hospitalization: | mITT Population |
| | | Kaplan-Meier plot, stratified by sex | · |
| | 14.2.2.6.18 | Time to first heart failure hospitalization: | mITT Population |
| | | Kaplan-Meier plot, stratified by heart failure | |
| | | ejection fraction | |
| | 14.2.2.6.19 | Time to first heart failure hospitalization: | Per Protocol |
| | | Kaplan-Meier plot | Population |
| | 14.2.2.6.20 | Time to first heart failure hospitalization: | Cohort #1 Population |
| | | Kaplan-Meier plot | |
| | 14.2.2.6.21 | Time to first heart failure emergency | mITT Population |
| | | department/hospital outpatient IV diuretic: | |
| | | Kaplan-Meier plot | |
| | 14.2.2.6.22 | Time to first heart failure emergency | mITT Population |
| | | department/hospital outpatient IV diuretic: | |
| | | Kaplan-Meier plot, stratified by sex | |
| | 14.2.2.6.23 | Time to first heart failure emergency | mITT Population |
| | | department/hospital outpatient IV diuretic: | |
| | | Kaplan-Meier plot, stratified by heart failure | |
| | | ejection fraction | |
| | 14.2.2.6.24 | Time to first heart failure emergency | Per Protocol |
| | | department/hospital outpatient IV diuretic: | Population |
| | | Kaplan-Meier plot | |
| | 14.2.2.6.25 | Time to first heart failure emergency | Cohort #1 Population |
| | | department/hospital outpatient IV diuretic: | |
| | | Kaplan-Meier plot | |
| | 14.2.2.6.41 | Time to first heart failure hospitalization from | mITT Population |
| | | CEC adjudication results: Kaplan-Meier plot | |
| | 14.2.2.6.42 | Time to first heart failure hospitalization from | mITT Population |
| | | CEC adjudication results: Kaplan-Meier plot, | |
| | 14400040 | stratified by sex | maITT Damid-4: |
| | 14.2.2.6.43 | Time to first heart failure hospitalization from | mITT Population |
| | | CEC adjudication results: Kaplan-Meier plot, | |
| | 14 2 2 6 44 | stratified by heart failure ejection fraction | Dor Drotocal |
| | 14.2.2.6.44 | Time to first heart failure hospitalization from | Per Protocol |
| | 1400045 | CEC adjudication results: Kaplan-Meier plot | Population |
| | 14.2.2.6.45 | Time to first heart failure hospitalization from | Cohort #1 Population |
| <u> </u> | 14 2 2 6 46 | CEC adjudication results: Kaplan-Meier plot | mITT Donutation |
| | 14.2.2.6.46 | Time to first heart failure emergency department/hospital outpatient IV diuretic from | mITT Population |
| | 14 2 2 6 47 | CEC adjudication results: Kaplan-Meier plot | mITT Donutation |
| | 14.2.2.6.47 | Time to first heart failure emergency department/hospital outpatient IV diuretic from | mITT Population |
| | | CEC adjudication results: Kaplan-Meier plot, | |
| | | stratified by sex | |
| | 1 | Straumed by Sex | |

| Header | Table Number | Name | Analysis Set |
|---|---|---|---|
| | 14.2.2.6.48 | Time to first heart failure emergency | mITT Population |
| | | department/hospital outpatient IV diuretic from | · |
| | | CEC adjudication results: Kaplan-Meier plot, | |
| | | stratified by heart failure ejection fraction | |
| | 14.2.2.6.49 | Time to first heart failure emergency | Per Protocol |
| | | department/hospital outpatient IV diuretic from | Population |
| | 1100000 | CEC adjudication results: Kaplan-Meier plot | |
| | 14.2.2.6.50 | Time to first heart failure emergency | Cohort #1 Population |
| | | department/hospital outpatient IV diuretic from | |
| | 140070 | CEC adjudication results: Kaplan-Meier plot | maITT Demulation |
| | 14.2.2.7.6 | Time to all-cause mortality: Kaplan-Meier plot | mITT Population |
| | 14.2.2.7.7 | Time to all-cause mortality: Kaplan-Meier plot, | mITT Population |
| | 14.2.2.7.8 | stratified by sex Time to all-cause mortality: Kaplan-Meier plot, | mITT Population |
| | 14.2.2.7.0 | stratified by heart failure ejection fraction | min i Population |
| | 14.2.2.7.9 | Time to all-cause mortality: Kaplan-Meier plot | Per Protocol |
| | 17.2.2.1.3 | Time to all-cause mortality. Napian-inciel plut | Population |
| | 14.2.2.7.10 | Time to all-cause mortality: Kaplan-Meier plot | Cohort #1 Population |
| | 14.2.2.7.11 | Time to cardiac mortality: Kaplan-Meier plot | mITT Population |
| | 14.2.2.7.12 | Time to cardiac mortality: Kaplan-Meier plot, | mITT Population |
| | | stratified by sex | I- 2 <del>.</del> |
| | 14.2.2.7.13 | Time to cardiac mortality: Kaplan-Meier plot, | mITT Population |
| | <u> </u> | stratified by heart failure ejection fraction | |
| | 14.2.2.7.14 | Time to cardiac mortality: Kaplan-Meier plot | Per Protocol |
| | | • | Population |
| | 14.2.2.7.15 | Time to cardiac mortality: Kaplan-Meier plot | Cohort #1 Population |
| | 14.2.2.7.21 | Time to all-cause mortality from CEC | mITT Population |
| | | adjudication results: Kaplan-Meier plot | |
| | 14.2.2.7.22 | Time to all-cause mortality from CEC | mITT Population |
| | | adjudication results: Kaplan-Meier plot, | |
| | 1100=00 | stratified by sex | |
| | 14.2.2.7.23 | Time to all-cause mortality from CEC | mITT Population |
| | | adjudication results: Kaplan-Meier plot, | |
| | 14.2.2.7.24 | stratified by heart failure ejection fraction | Dor Drotocal |
| | 14.2.2.1.24 | Time to all-cause mortality from CEC | Per Protocol |
| | 14.2.2.7.25 | adjudication results: Kaplan-Meier plot Time to all-cause mortality from CEC | Population Cohort #1 Population |
| | 14.2.2.7.20 | adjudication results: Kaplan-Meier plot | Conon #1 Population |
| | 14.2.2.7.26 | Time to cardiac mortality from CEC | mITT Population |
| | 17.2.2.1.20 | adjudication results: Kaplan-Meier plot | min i opulation |
| | 14.2.2.7.27 | Time to cardiac mortality from CEC | mITT Population |
| | | adjudication results: Kaplan-Meier plot, | I- 2 <del>.</del> |
| | | stratified by sex | |
| | 14.2.2.7.28 | Time to cardiac mortality from CEC | mITT Population |
| | | adjudication results: Kaplan-Meier plot, | ' |
| | | stratified by heart failure ejection fraction | |
| | 14.2.2.7.29 | Time to cardiac mortality from CEC | Per Protocol |
| | | adjudication results: Kaplan-Meier plot | Population |
| | 14.2.2.7.30 | Time to cardiac mortality from CEC | Cohort #1 Population |
| | | adjudication results: Kaplan-Meier plot | |
| 14.3 | | Safety Data Summary Figures and Tables | |
| 14.3.1.1 | | Primary Safety Endpoint | |

| Header Table Number | | Name | Analysis Set |
|---|---|---|---|
| | 14.3.1.1.8 | Freedom from device/system related | mITT Population |
| | | complication: Kaplan-Meier plot | |
| | 14.3.1.1.9 | Freedom from device/system related | mITT Population |
| | | complication: Kaplan-Meier plot, stratified by | |
| | | sex | |
| | 14.3.1.1.10 | Freedom from device/system related | mITT Population |
| | | complication: Kaplan-Meier plot, stratified by | |
| | | heart failure ejection fraction | |
| | 14.3.1.1.11.1 | Freedom from device/system related | Per Protocol |
| | 4404440 | complication : Kaplan-Meier plot | Population |
| | 14.3.1.1.11.2 | Freedom from device/system related | ITT Population |
| | 4404440 | complication : Kaplan-Meier plot | O-1 |
| | 14.3.1.1.12 | Freedom from device/system related | Cohort #1 Population |
| | 4404400 | complication : Kaplan-Meier plot | ITT Danielettan |
| | 14.3.1.1.20 | Freedom from device/system related | mITT Population |
| | | complication from CEC adjudication results:<br>Kaplan-Meier plot | |
| | 14.3.1.1.21 | Freedom from device/system related | mITT Population |
| | 14.3.1.1.21 | complication from CEC adjudication results: | IIII I Fopulation |
| | | Kaplan-Meier plot, stratified by sex | |
| | 14.3.1.1.22 | Freedom from device/system related | mITT Population |
| | 14.5.1.1.22 | complication from CEC adjudication results: | IIII I I Opulation |
| | | Kaplan-Meier plot, stratified by heart failure | |
| | | ejection fraction | |
| | 14.3.1.1.23.1 | Freedom from device/system related | Per Protocol |
| | | complication from CEC adjudication results: | Population |
| | | Kaplan-Meier plot | ' |
| | 14.3.1.1.23.2 | Freedom from device/system related | ITT Population |
| | | complication from CEC adjudication results: | |
| | | Kaplan-Meier plot | |
| | 14.3.1.1.24 | Freedom from device/system related | Cohort #1 Population |
| | | complication from CEC adjudication results: | |
| | 110100 | Kaplan-Meier plot | |
| | 14.3.1.2.8 | Freedom from pressure sensor failure: | mITT Population |
| | 440400 | Kaplan-Meier plot | |
| | 14.3.1.2.9 | Freedom from pressure sensor failure: | mITT Population |
| | 1424240 | Kaplan-Meier plot, stratified by sex | mITT Donutation |
| | 14.3.1.2.10 | Freedom from pressure sensor failure: | mITT Population |
| | | Kaplan-Meier plot, stratified by heart failure ejection fraction | |
| | 14.3.1.2.11.1 | Freedom from pressure sensor failure: | Per Protocol |
| | 14.5.1.2.11.1 | Kaplan-Meier plot | Population |
| | 14.3.1.2.11.2 | Freedom from pressure sensor failure: | ITT Population |
| | 17.0.1.2.11.2 | Kaplan-Meier plot | TITT Opulation |
| | 14.3.1.2.12 | Freedom from pressure sensor failure: | Cohort #1 Population |
| | 17.0.1.2.12 | Kaplan-Meier plot | Conort // 1 opulation |
| | 14.3.1.2.20 | Freedom from pressure sensor failure from | mITT Population |
| | | CEC adjudication results: Kaplan-Meier plot | |
| | 14.3.1.2.21 | Freedom from pressure sensor failure from | mITT Population |
| | | CEC adjudication results: Kaplan-Meier plot, | ' |
| | | stratified by sex | |

| Header | Table Number | Name | Analysis Set |
|---|---|---|---|
| | 14.3.1.2.22 | Freedom from pressure sensor failure from CEC adjudication results: Kaplan-Meier plot, stratified by heart failure ejection fraction | mITT Population |
| | 14.3.1.2.23.1 | Freedom from pressure sensor failure from | Per Protocol |
| | | CEC adjudication results: Kaplan-Meier plot | Population |
| | 14.3.1.2.23.2 | Freedom from pressure sensor failure from CEC adjudication results: Kaplan-Meier plot | ITT Population |
| | 14.3.1.2.24 | Freedom from pressure sensor failure from CEC adjudication results: Kaplan-Meier plot | Cohort #1 Population |

# 16. Index of Listings

| Header | Table Number | Name | Analysis Set |
|---|---|---|---|
| 16.2 | | Subject Data Listings | |
| 16.2.1 | | Discontinued Subjects | |
| | 16.2.1.1.1 | Subject disposition, part 1 | Enrolled Population |
| | 16.2.1.1.1.1 | Subject disposition, part 1 | Cohort #1 |
| | | | Population |
| | 16.2.1.1.2 | Subject disposition, part 2 | Enrolled Population |
| | 16.2.1.1.2.1 | Subject disposition, part 2 | Cohort #1 |
| | | | Population |
| | 16.2.1.2 | Eligibility safety approval provided by Eligibility committee (EC) | Enrolled Population |
| | 16.2.1.2.1 | Eligibility safety approval provided by | Cohort #1 |
| | 16.2.1.3 | Eligibility committee (EC) Subject status | Population Enrolled Population |
| | 16.2.1.3.1 | Subject status | Cohort #1<br>Population |
| | 16.2.1.4 | Subject training at implant visit | Enrolled Population |
| | 16.2.1.4.1 | Subject training at implant visit | Cohort #1 |
| | | | Population |
| 16.2.2 | | Protocol Deviations | |
| | 16.2.2.1 | Protocol deviations and non-<br>compliance | Enrolled Population |
| | 16.2.2.1.1 | Protocol deviations and non- | Cohort #1 |
| | | compliance | Population |
| 16.2.3 | | Subjects Excluded from the Efficacy Analysis | |
| | 16.2.3.1 | Inclusion criteria | |
| | 16.2.3.2 | Exclusion criteria | |
| | 16.2.3.3 | Exclusions from analysis sets | Enrolled Population |
| | 16.2.3.4 | Screen failures and primary reason for screen failure | Screen Failure |
| 16.2.4 | | Demographic Data | |
| | 16.2.4.1 | Demographics | Enrolled Population |
| | 16.2.4.1.1 | Demographics | Cohort #1 |
| | | | Population |
| | 16.2.4.2 | Medical history | Enrolled Population |
| | 16.2.4.2.1 | Medical history | Cohort #1 |
| | | • | Population |
| | 16.2.4.3.1 | Cardiovascular history - general | Enrolled Population |
| | 16.2.4.3.1.1 | Cardiovascular history - general | Cohort #1 |
| | | | Population |
| | 16.2.4.3.2 | Cardiovascular history – past year | Enrolled Population |
| | 16.2.4.3.2.1 | Cardiovascular history – past year | Cohort #1 Population |
| | 16.2.4.4 | Cardiac medical and surgical history | Enrolled Population |
| | 16.2.4.4.1 | Cardiac medical and surgical history | Cohort #1<br>Population |
| | 16.2.4.5 | Baseline and concomitant medications | Enrolled Population |

This document is confidential.

SAP Version: 3.0 dated 17-Aug-2023 Controlled Document ID: **3903A.01**, Effective Date 29-Oct-2018

| Header | Table Number | Name | Analysis Set |
|---|---|---|---|
| | 16.2.4.5.1 | Baseline and concomitant | Cohort #1 |
| | | medications | Population |
| 16.2.5 | | System Use Compliance – Not | |
| | | applicable | |
| 16.2.6 | | Individual Efficacy Data | |
| | 16.2.6.1 | Cordella sensor implant | Enrolled Population |
| | 16.2.6.2 | Mortality | Enrolled Population |
| | 16.2.6.2.1 | Mortality | Cohort #1 |
| | | | Population |
| | 16.2.6.3 | Hospitalization | Enrolled Population |
| | 16.2.6.3.1 | Hospitalization | Cohort #1 |
| | | · | Population |
| | 16.2.6.4 | Emergency department/hospital | Enrolled Population |
| | | outpatient IV diuretic visits | |
| | 16.2.6.4.1 | Emergency department/hospital | Cohort #1 |
| | | outpatient IV diuretic visits | Population |
| | 16.2.6.5 | Heart failure related medication | Enrolled Population |
| | | changes | · |
| | 16.2.6.5.1 | Heart failure related medication | Cohort #1 |
| | | changes | Population |
| | 16.2.6.6 | Cordella sensor PAP measurements | Enrolled Population |
| | 16.2.6.7 | Quality of life KCCQ questionnaire | Enrolled Population |
| | 16.2.6.7.1 | Quality of life KCCQ questionnaire | Cohort #1 |
| | 10.2.0.7.1 | addity of inc 1000 quodiofinanc | Population |
| | 16.2.6.8 | NYHA functional classification | Enrolled Population |
| | 16.2.6.8.1 | NYHA functional classification | Cohort #1 |
| | 10.2.0.0.1 | TTT W T another an elacenteation | Population |
| | 16.2.6.9 | Six (6) minute walk test | Enrolled Population |
| | 16.2.6.9.1 | Six (6) minute walk test | Cohort #1 |
| | 10.2.0.0.1 | Oix (o) minute want toot | Population |
| | 16.2.6.10 | RHC PAP measurements | Enrolled Population |
| | 16.2.6.10.1 | RHC PAP measurements | Cohort #1 |
| | 10.2.0.10.1 | Tale 17 a measurements | Population |
| 16.2.7 | | Adverse Event Listings | · |
| | 16.2.7.1 | Adverse events | Enrolled Population |
| | 16.2.7.1.1 | Adverse events | Cohort #1 |
| | | | Population |
| | 16.2.7.2 | Device/system related complications | Enrolled Population |
| | 16.2.7.2.1 | Device/system related complications | Cohort #1 |
| | | , , | Population |
| | 16.2.7.3 | Device Deficiency | Enrolled Population |
| | 16.2.7.3.1 | Device Deficiency | Cohort #1 |
| | | | Population |
| | 16.2.7.4 | Predefined adverse events by | Enrolled Population |
| | | category adjudicated by CEC | <u>'</u> |
| | 16.2.7.4.1 | Predefined adverse events by | Cohort #1 |
| | | category adjudicated by CEC | Population |
| | 16.2.7.5 | CEC adjudication results | Enrolled Population |
| | 16.2.7.5.1 | CEC adjudication results | Cohort #1 |
| | | | Population |
| | | | ι υραιατίστι |

| Header | Table Number | Name | Analysis Set |
|---|---|---|---|
| 16.2.8 | | Listing of individual laboratory | |
| | | measurements by subject | |
| | 16.2.8.1 | Clinical Laboratory Data | |
| | 16.2.8.1.1 | Hematology | Enrolled Population |
| | 16.2.8.1.1.1 | Hematology | Cohort #1 |
| | | | Population |
| | 16.2.8.1.2 | Chemistry | Enrolled Population |
| | 16.2.8.1.2.1 | Chemistry | Cohort #1 |
| | | | Population |
| | 16.2.8.1.3 | Urinalysis | Enrolled Population |
| | 16.2.8.1.3.1 | Urinalysis | Cohort #1 |
| | | | Population |
| | 16.2.8.1.4 | Coagulation | Enrolled Population |
| | 16.2.8.1.4.1 | Coagulation | Cohort #1 |
| | | | Population |
| | 16.2.8.1.5 | NT-pro BNP | Enrolled Population |
| | 16.2.8.1.5.1 | NT-pro BNP | Cohort #1 |
| | | | Population |
| | 16.2.8.1.6 | Pregnancy test | Enrolled Population |
| | 16.2.8.1.6.1 | Pregnancy test | Cohort #1 |
| | | | Population |
| | 16.2.8.2 | Other Safety Data | |
| | 16.2.8.2.1 | Vital signs | Enrolled Population |
| | 16.2.8.2.1.1 | Vital signs | Cohort #1 |
| | | | Population |
| | 16.2.8.2.2 | Electrocardiogram (ECG) | Enrolled Population |
| | 16.2.8.2.2.1 | Electrocardiogram (ECG) | Cohort #1 |
| | | | Population |
| | 16.2.8.2.3 | Echocardiogram | Enrolled Population |
| | 16.2.8.2.3.1 | Echocardiogram | Cohort #1 |
| | | | Population |
| | 16.2.8.2.4 | Physical Examination | Enrolled Population |
| | 16.2.8.2.4.1 | Physical Examination | Cohort #1 |
| | | | Population |

# 17. Appendices

This document is confidential.

SAP Version: 3.0 dated 17-Aug-2023 Controlled Document ID: **3903A.01**, Effective Date 29-Oct-2018 Filing requirements: TMF

#### 17.1. Appendix 1: Time and Event Schedule

| Assessment | V1:<br>Screening/<br>Enrollment<br>(30 days) <sup>15</sup> | V2:<br>Cordella PA<br>Sensor<br>Implant Visit | V3:<br>Month<br>1<br>(±7 days) | V4 <sup>11</sup> :<br>Month<br>3<br>(±7 days) | V5:<br>Month<br>6<br>(±14 days) | V6:<br>Month<br>12<br>(±30 days) | V7 to V8:<br>Months 18,<br>24<br>(±30 days) | V9 to V11<br>Year<br>3, 4, 5<br>(±30 days) |
|---|---|---|---|---|---|---|---|---|
| Informed Consent | Х | | | | | | | |
| Subject Demographics | Х | | | | | | | |
| Study Eligibility Review and Committee Approval | Х | | | | | | | |
| Cardiac/Medical & Surgical History | Х | | | | | | | |
| Physical Exam, height, weight, and vital signs <sup>1, 5</sup> | Х | Х | X <sup>12</sup> | | Х | Х | Х | Х |
| 12-Lead ECG with Interpretation | Х | | | | Х | Х | X <sup>4</sup> | X |
| Urinalysis <sup>2</sup> | Х | | | | | | | |
| Safety Labs (Chemistry/Hematology/ aPTT/ INR) | Х | | | | Х | Х | X <sup>4</sup> | Х |
| Serum NT-pro BNP | Х | | Х | X <sup>12</sup> | Х | Х | Х | X |
| aPTT/ INR (if indicated) | | | | | | | | |
| Echocardiogram <sup>3</sup> | Х | | | | | Х | | Х |
| Subject Training: Cordella™ HF System <sup>14</sup> | Х | | | | | | | |
| Subject Training: CorPASS | | X | | | | | | |
| Cordella™ PA Sensor Implant | | Х | | | | | | |
| Cordella System Use (daily) | Х | X | Х | Х | Х | X | Х | Х |
| Cordella™ PAP – dia/sys/mean/pulse | | X <sub>9</sub> | X <sup>5,6</sup> | X <sup>5,6</sup> | X <sup>5,6</sup> | X <sup>5,6</sup> | X <sup>5,6</sup> | X <sub>6</sub> |
| RHC PAP / RAP/ PCWP/ CO/ CI/ RVP8 | | Х | | | | | | X <sup>12</sup> |
| Subject Status | Х | | Х | Х | X <sup>10</sup> | X <sup>10</sup> | Х | X |
| 6- Minute Walk Test | Х | | | | Х | X <sup>7</sup> | X <sup>4,7</sup> | X <sup>7</sup> |
| NYHA Functional Classification | X <sup>16</sup> | | Х | Х | Х | Х | Х | Х |
| KCCQ Quality of Life Questionnaires 5 | Х | | Х | Х | Х | Х | Х | Х |
| Concurrent/Cardiac Medications | Х | Х | Х | Х | Х | Х | Х | Х |
| Adverse Events | Х | Х | Х | Х | Х | Х | Х | Х |
| Health Economic Questionnaire | | | | | | | X <sup>4</sup> | |
| Subject Survey (optional)/ Cohort #1 only 13 | Month 1 after Unblinding Quarterly until V11 / Year 5 | | | | | | | |
| Site Survey (optional)/ Cohort #1 only <sup>13</sup> | <ul><li>1. Month 1 after Unblinding</li><li>2. Quarterly until V11 / Year 5</li></ul> | | | | | | | |
| Full Physical Examination and Height performed at Screening V Urine (V1) pregnancy test for females | isit only | | 8. Additional R<br>9. Via CalEQ | RHC as needed for | or Re-calibration p | ourposes at the cli | nician's discretion | |

This document is confidential.


Controlled Document ID: 3903A.01, Effective Date 29-Oct-2018

Sponsor: Endotronix, Protocol No.: ETX-HFS-PA-03

- 3. Echo may be obtained within 3 or 6 months of Screening details are in protocol section 8.1.10
- 4. At Month 24 only
- 5. via myCordella™ Patient App at home prior to visit. Baseline KCCQ will be completed on myCordella tablet following Cordella System distribution at Screening Visit
- 6. via myCordella™ Patient App sitting and supine
- 7. Additional PAP Measurements will be obtained before and after 6-minute walk test

- 10. Incl. question on assigned treatment at Visit 5 and 6
- 11. Visit should be completed remote/virtually
- 12. If available
- 13. After subject gets unblinded to PAP Pressures at V6 or cross-over whatever comes first
- 14. Subject training on and distribution of the commercial Cordella™ System (should occur at Screening Visit (Visit 1).
- 15. Some study procedures need to be repeated in case a subject is implanted >30 days after Visit 1, details are in protocol section 8.3.1
- 16. may be obtained within the 30 day Study Visit 1 window
- 17. At V9 / Year 3 only

#### 17.2. Appendix 2: The Kansas City Cardiomyopathy Questionnaire Scoring Instructions

Note: references to "means of questions actually answered" imply the following.

If there are n questions in a scale, and the subject must answer m to score the scale, but the subject answers only n-i, where n-i >= m, calculate the **mean of those questions** as (sum of the responses to those n-i questions) / (n-i)

not

(sum of the responses to those *n-i* questions) / *n* 

There are 10 summary scores within the KCCQ, which are calculated as follows:

#### 1. Physical Limitation

Code responses to each of Questions 1a-f as follows:

Extremely limited = 1

Quite a bit limited = 2

Moderately limited = 3

Slightly limited = 4

Not at all limited = 5

Limited for other reasons or did not do = <missing value>

If at least three of Questions 1a-f are not missing, then compute

Physical Limitation Score = 100\*[(mean of Questions 1a-f actually answered) – 1]/4

#### 2. Symptom Stability

•Code the response to Question 2 as follows:

This document is confidential.


Controlled Document ID: 3903A.01, Effective Date 29-Oct-2018

Much worse = 1

Slightly worse = 2

Not changed = 3

Slightly better = 4

Much better = 5

I've had no symptoms over the last 2 weeks = 3

If Question 2 is not missing, then compute

Symptom Stability Score = 100\*[(Question 2) - 1]/4

#### 3. Symptom Frequency

Code responses to Questions 3, 5, 7 and 9 as follows:

#### Question 3

Every morning = 1

3 or more times a week but not every day = 2

1-2 times a week = 3

Less than once a week = 4

Never over the past 2 weeks = 5

#### Questions 5 and 7

All of the time = 1

Several times a day = 2

At least once a day = 3

3 or more times a week but not every day = 4

1-2 times a week = 5

Less than once a week = 6

Never over the past 2 weeks = 7

#### Question 9

Every night = 1

This document is confidential.

3 or more times a week but not every day = 2

1-2 times a week = 3

Less than once a week = 4

Never over the past 2 weeks = 5

If at least two of Questions 3, 5, 7 and 9 are not missing, then compute:

S3 = [(Question 3) - 1]/4

S5 = [(Question 5) - 1]/6

S7 = [(Question 7) - 1]/6

S9 = [(Question 9) - 1]/4

Symptom Frequency Score = 100\*(mean of S3, S5, S7 and S9)

#### 4. Symptom Burden

Code responses to each of Questions 4, 6 and 8 as follows:

Extremely bothersome = 1

Quite a bit bothersome = 2

Moderately bothersome = 3

Slightly bothersome = 4

Not at all bothersome = 5

I've had no swelling/fatigue/shortness of breath = 5

If at least one of Questions 4, 6 and 8 is not missing, then compute Symptom Burden Score = 100\*[(mean of Questions 4, 6 and 8 actually answered) – 1]/4

#### 5. Total Symptom Score

= mean of the following available summary scores: Symptom Frequency Score and Symptom Burden Score

#### 6. Self-Efficacy

Code responses to Questions 10 and 11 as follows:

#### Question 10

Not at all sure = 1

Not very sure = 2

Somewhat sure = 3

This document is confidential.


Controlled Document ID: 3903A.01, Effective Date 29-Oct-2018

Mostly sure = 4

Completely sure = 5

#### Question 11

Do not understand at all = 1

Do not understand very well = 2

Somewhat understand = 3

Mostly understand = 4

Completely understand = 5

If at least one of Questions 10 and 11 is not missing, then compute Self-Efficacy Score = 100\*[(mean of Questions 10 and 11 actually answered) – 1]/4

#### 7. Quality of Life

#### Code responses to Questions 12, 13 and 14 as follows:

#### Question 12

It has extremely limited my enjoyment of life = 1

It has limited my enjoyment of life quite a bit = 2

It has moderately limited my enjoyment of life = 3

It has slightly limited my enjoyment of life = 4

It has not limited my enjoyment of life at all = 5

#### Question 13

Not at all satisfied = 1

Mostly dissatisfied = 2

Somewhat satisfied = 3

Mostly satisfied = 4

Completely satisfied = 5

#### Question 14

I felt that way all of the time = 1

This document is confidential.


Controlled Document ID: 3903A.01, Effective Date 29-Oct-2018

Sponsor: Endotronix, Protocol No.: ETX-HFS-PA-03

I felt that way most of the time = 2

I occasionally felt that way = 3

I rarely felt that way = 4

I never felt that way = 5

If at least one of Questions 12, 13 and 14 is not missing, then compute Quality of Life Score = 100\*[(mean of Questions 12, 13 and 14 actually answered) – 1]/4

#### 8. Social Limitation

Code responses to each of Questions 15a-d as follows:

Severely limited = 1

Limited quite a bit = 2

Moderately limited = 3

Slightly limited = 4

Did not limit at all = 5

Does not apply or did not do for other reasons = <missing value>

If at least two of Questions 15a-d are not missing, then compute

Social Limitation Score = 100\*[(mean of Questions 15a-d actually answered) – 1]/4

#### 9. Overall Summary Score

= mean of the following available summary scores: Physical Limitation Score, Total Symptom Score, Quality of Life Score, Social Limitation Score

#### 10. Clinical Summary Score

= mean of the following available summary scores: Physical Limitation Score, Total Symptom Score

# 7000235\_Statistical Analysis Plan\_v3.0\_17Aug2023

Final Audit Report 2023-08-17

Created: 2023-08-17

By: Stone Liu (stone.liu@syneoshealth.com)

Status: Signed

Transaction ID: CBJCHBCAABAAIO7BqNBc8C6a4r3Y150LLHHt04JFU09L

# "7000235\_Statistical Analysis Plan\_v3.0\_17Aug2023" History

- Document created by stone.liu@syneoshealth.com 2023-08-17 6:56:29 AM GMT
- Document emailed to stone.liu@syneoshealth.com for signature 2023-08-17 6:57:43 AM GMT
- Document emailed to tianzhe.liu@syneoshealth.com for signature 2023-08-17 6:57:44 AM GMT
- Document emailed to wesley.basson@syneoshealth.com for signature 2023-08-17 6:57:44 AM GMT
- Document emailed to Andrea Sauerland (andrea.sauerland@endotronix.com) for signature 2023-08-17 6:57:44 AM GMT
- Signer stone.liu@syneoshealth.com entered name at signing as Stone Liu 2023-08-17 6:58:42 AM GMT
- Stone Liu (stone.liu@syneoshealth.com) authenticated with Adobe Acrobat Sign. 2023-08-17 6:58:44 AM GMT
- Document e-signed by Stone Liu (stone.liu@syneoshealth.com)

Signing reason: I am the author

Signature Date: 2023-08-17 - 6:58:44 AM GMT - Time Source: server

- Email viewed by Andrea Sauerland (andrea.sauerland@endotronix.com) 2023-08-17 7:09:03 AM GMT
- Andrea Sauerland (andrea.sauerland@endotronix.com) authenticated with Adobe Acrobat Sign. 2023-08-17 - 7:11:17 AM GMT





Document e-signed by Andrea Sauerland (andrea.sauerland@endotronix.com)

Signing reason: I am the approver

Signature Date: 2023-08-17 - 7:11:17 AM GMT - Time Source: server

Email viewed by wesley.basson@syneoshealth.com

2023-08-17 - 8:27:12 AM GMT

Signer wesley.basson@syneoshealth.com entered name at signing as Wesley Basson 2023-08-17 - 8:28:49 AM GMT

Wesley Basson (wesley.basson@syneoshealth.com) authenticated with Adobe Acrobat Sign. 2023-08-17 - 8:28:51 AM GMT

Document e-signed by Wesley Basson (wesley.basson@syneoshealth.com)

Signing reason: I am the approver

Signature Date: 2023-08-17 - 8:28:51 AM GMT - Time Source: server

Signer tianzhe.liu@syneoshealth.com entered name at signing as Tianzhe Liu 2023-08-17 - 9:52:49 AM GMT

✓ Tianzhe Liu (tianzhe.liu@syneoshealth.com) authenticated with Adobe Acrobat Sign. 2023-08-17 - 9:52:51 AM GMT

Document e-signed by Tianzhe Liu (tianzhe.liu@syneoshealth.com)

Signing reason: I am the reviewer

Signature Date: 2023-08-17 - 9:52:51 AM GMT - Time Source: server

Agreement completed.

2023-08-17 - 9:52:51 AM GMT

